CLINICAL TRIAL: NCT02484690
Title: A Multiple-Center, Multiple-Dose and Regimen, Randomized, Active Comparator Controlled, Double-Masked, Parallel Group, 36 Week Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Efficacy of RO6867461 Administered Intravitreally in Patients With Choroidal Neovascularization Secondary to Age-Related Macular Degeneration
Brief Title: A Proof-of-Concept Study of Faricimab (RO6867461) in Participants With Choroidal Neovascularization (CNV) Secondary to Age-Related Macular Degeneration (AMD)
Acronym: AVENUE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BP29647
Record Dates: First submitted 2015-06-12; First posted 2015-06-30 (Estimated); Results first posted 2020-10-09 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-10

CONDITIONS: Choroidal Neovascularization
MeSH Terms: conditions — Choroidal Neovascularization | interventions — faricimab; Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) (Active Comparator): Participants will receive ranibizumab, 0.5 milligrams (mg) intravitreal (IVT) Q4W up to Week 32 (total 9 injections). The final study visit will take place at Week 36.
  Interventions: Drug: Ranibizumab
- Arm B: Faricimab, 1.5 mg Q4W (Experimental): Participants will receive faricimab 1.5 mg IVT Q4W up to Week 32 (total 9 injections). The final study visit will take place at Week 36.
  Interventions: Drug: Faricimab
- Arm C: Faricimab, 6 mg Q4W (Experimental): Participants will receive faricimab 6 mg IVT Q4W up to Week 32 (9 injections). The final study visit will take place at Week 36.
  Interventions: Drug: Faricimab
- Arm D: Faricimab, 6 mg Every 4-8 weeks (Experimental): Participants will receive faricimab, 6 mg IVT Q4W up to Week 12 (4 injections), followed by 6 mg IVT every 8 weeks up to Week 28 (2 injections). On Weeks 16, 24, and 32, participants received the sham procedure in order to maintain masking. The final study visit will take place at Week 36.
  Interventions: Drug: Faricimab; Drug: Sham Procedure
- Arm E: Ranibizumab 0.5 mg + Faricimab 6 mg Q4W (Experimental): Participants will receive ranibizumab, 0.5 mg IVT Q4W up to Week 8 (3 injections), followed by faricimab, 6 mg IVT Q4W up to Week 32 (6 injections). The final study visit will take place at Week 36.
  Interventions: Drug: Faricimab; Drug: Ranibizumab

INTERVENTIONS:
Drug: Faricimab — Faricimab will be administered as per the regimen specified in the individual arm.
  Other Names: RO6867461; RG7716
  Arms: Arm B: Faricimab, 1.5 mg Q4W; Arm C: Faricimab, 6 mg Q4W; Arm D: Faricimab, 6 mg Every 4-8 weeks; Arm E: Ranibizumab 0.5 mg + Faricimab 6 mg Q4W
Drug: Ranibizumab — Ranibizumab will be administered as per the regimen specified in the individual arm.
  Other Names: Lucentis
  Arms: Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W); Arm E: Ranibizumab 0.5 mg + Faricimab 6 mg Q4W
Drug: Sham Procedure — The sham is a procedure that mimics an intravitreal injection, but involves the blunt end of an empty syringe (without a needle) being pressed against the anesthetized eye. It will be administered to participants in treatment arm D at applicable visits to maintain masking.
  Arms: Arm D: Faricimab, 6 mg Every 4-8 weeks

SUMMARY:
This multiple-center, multiple-dose and regimen, randomized, double-masked active comparator-controlled, double-masked, five parallel group, 36-week study will evaluate the efficacy, safety, tolerability, and pharmacokinetics of faricimab (RO6867461) in participants with choroidal neovascularization (CNV) secondary to age-related macular degeneration (AMD).

The study was designed to allow the evaluation of RO6867461 in a treatment-naive population (comparison of Arms A, B, C, and D) and an anti-VEGF-incomplete responder population that met a predefined criterion at Week 12 (comparison between Arms A and E). Only one eye per participant was chosen as the study eye.

ELIGIBILITY:
Inclusion Criteria:

* Treatment-naive with CNV secondary to AMD, with subfoveal CNV or juxtafoveal CNV with a subfoveal component related to the CNV activity by FFA or SD-OCT
* Active CNV

Exclusion Criteria:

* CNV due to causes other than AMD
* Subretinal hemorrhage, fibrosis, or atrophy involving either the fovea or more than 50% of the total lesion area
* Cataract surgery within 3 months of baseline, or any other previous intraocular surgery
* Major illness or surgery within 1 month prior to Screening
* Glycosylated hemoglobin (HbA1c) above 7.5%
* Uncontrolled blood pressure

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 2015-08-11 (Actual); Primary Completion 2017-09-26 (Actual); Study Completion 2017-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (52):
- United States (52):
  - Associated Retina Consultants, Phoenix, Arizona
  - Retinal Consultants of Arizona, Phoenix, Arizona
  - California Retina Consultants, Bakersfield, California
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - The Retina Partners, Encino, California
  - Retina Consultants, San Diego, Poway, California
  - Orange County Retina Med Group, Santa Ana, California
  - Bay Area Retina Associates, Walnut Creek, California
  - American Institute of Research, Whittier, California
  - Retina Consultants of Southern, Colorado Springs, Colorado
  - Colorado Retina Associates, PC, Golden, Colorado
  - New England Retina Associates, Hamden, Connecticut
  - Retina Health Center, Fort Myers, Florida
  - National Ophthalmic Research Institute, Fort Myers, Florida
  - Florida Eye Associates, Melbourne, Florida
  - Central Florida Retina, Orlando, Florida
  - Retina Care Specialists, Palm Beach Gardens, Florida
  - Retina Vitreous Assoc of FL, St. Petersburg, Florida
  - Southern Vitreoretinal Assoc, Tallahassee, Florida
  - Southeast Retina Center, Augusta, Georgia
  - Georgia Retina PC, Marietta, Georgia
  - Midwest Eye Institute Northside, Indianapolis, Indiana
  - Paducah Retinal Center, Paducah, Kentucky
  - Retina Group of Washington, Chevy Chase, Maryland
  - National Retina Institute, Towson, Maryland
  - Vitreo-Retinal Associates, PC, Worcester, Massachusetts
  - Vitreoretinal Surgery, Edina, Minnesota
  - Retina Associates of NJ, Toms River, New Jersey
  - Eye Associates of New Mexico, Albuquerque, New Mexico
  - Long Is. Vitreoretinal Consult, Great Neck, New York
  - Opthalmic Consultants of LI, Lynbrook, New York
  - Retina Assoc of Western NY, Rochester, New York
  - The Retina Consultants, Slingerlands, New York
  - Western Carolina Retinal Associate PA, Asheville, North Carolina
  - Char Eye Ear &Throat Assoc, Charlotte, North Carolina
  - OSU Eye Physicians & Surgeons, Columbus, Ohio
  - Oregon Retina, LLP, Eugene, Oregon
  - Oregon Retina institute, Medford, Oregon
  - Retina Northwest, Portland, Oregon
  - Mid Atlantic Retina, Philadelphia, Pennsylvania
  - Palmetto Retina Center, West Columbia, South Carolina
  - Southeastern Retina Associates Chattanooga, Chattanooga, Tennessee
  - Charles Retina Institute, Germantown, Tennessee
  - Tennessee Retina PC., Nashville, Tennessee
  - W Texas Retina Consultants PA, Abilene, Texas
  - Austin Retina Associates, Austin, Texas
  - Retina Research Center, Austin, Texas
  - Retina Consultants of Houston, Houston, Texas
  - Strategic Clinical Research Group, LLC, Willow Park, Texas
  - Retina Associates of Utah, Salt Lake City, Utah
  - Univ of Virginia Ophthalmology, Charlottesville, Virginia
  - Spokane Eye Clinical Research, Spokane, Washington

REFERENCES:
- [Derived] Kikuchi Y, Kawczynski MG, Anegondi N, Neubert A, Dai J, Ferrara D, Quezada-Ruiz C. Machine Learning to Predict Faricimab Treatment Outcome in Neovascular Age-Related Macular Degeneration. Ophthalmol Sci. 2023 Aug 18;4(2):100385. doi: 10.1016/j.xops.2023.100385. eCollection 2024 Mar-Apr. PMID 37868796
- [Derived] Yu S, Bachmeier I, Hernandez-Sanchez J, Garcia Armendariz B, Ebneter A, Pauleikhoff D, Chakravarthy U, Fauser S. Hyperreflective Material Boundary Remodeling in Neovascular Age-Related Macular Degeneration: A Post Hoc Analysis of the AVENUE Trial. Ophthalmol Retina. 2023 Nov;7(11):990-998. doi: 10.1016/j.oret.2023.06.024. Epub 2023 Jul 6. PMID 37422192
- [Derived] Maunz A, Benmansour F, Li Y, Albrecht T, Zhang YP, Arcadu F, Zheng Y, Madhusudhan S, Sahni J. Accuracy of a Machine-Learning Algorithm for Detecting and Classifying Choroidal Neovascularization on Spectral-Domain Optical Coherence Tomography. J Pers Med. 2021 Jun 8;11(6):524. doi: 10.3390/jpm11060524. PMID 34201045
- [Derived] Sahni J, Dugel PU, Patel SS, Chittum ME, Berger B, Del Valle Rubido M, Sadikhov S, Szczesny P, Schwab D, Nogoceke E, Weikert R, Fauser S. Safety and Efficacy of Different Doses and Regimens of Faricimab vs Ranibizumab in Neovascular Age-Related Macular Degeneration: The AVENUE Phase 2 Randomized Clinical Trial. JAMA Ophthalmol. 2020 Sep 1;138(9):955-963. doi: 10.1001/jamaophthalmol.2020.2685. PMID 32729888

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 273 patients were randomized, but 10 participants in total were excluded from the analysis populations, 1, 3, 1, and 5 from Arms B, C, D, and E, respectively, because of Good Clinical Practice (GCP) violations at a single site.
Groups:
- Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W): Participants received ranibizumab, 0.5 milligrams (mg) intravitreal (IVT) once every 4 weeks (Q4W) up to Week 32 (total 9 injections). The final study visit took place at Week 36.
- Arm B: Faricimab, 1.5 mg Q4W: Participants received faricimab 1.5 mg IVT Q4W up to Week 32 (total 9 injections). The final study visit took place at Week 36.
- Arm C: Faricimab, 6 mg Q4W: Participants received faricimab 6 mg IVT Q4W up to Week 32 (9 injections). The final study visit took place at Week 36.
- Arm D: Faricimab, 6 mg Every 4-8 Weeks: Participants received faricimab, 6 mg IVT Q4W up to Week 12 (4 injections), followed by 6 mg IVT every 8 weeks up to Week 28 (2 injections). On Weeks 16, 24, and 32, participants received the sham procedure in order to maintain masking. The final study visit took place at Week 36.
- Arm E: Ranibizumab 0.5 mg + Faricimab 6 mg Q4W: Participants received ranibizumab, 0.5 mg IVT Q4W up to Week 8 (3 injections), followed by faricimab, 6 mg IVT Q4W up to Week 32 (6 injections). The final study visit took place at Week 36.
Period: Overall Study
Arm/Group | Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) | Arm B: Faricimab, 1.5 mg Q4W | Arm C: Faricimab, 6 mg Q4W | Arm D: Faricimab, 6 mg Every 4-8 Weeks | Arm E: Ranibizumab 0.5 mg + Faricimab 6 mg Q4W
Started | 68 | 46 | 39 | 46 | 64
Received at Least One Dose of Study Drug (Safety Population) | 67 | 46 | 39 | 46 | 64
Completed | 64 | 40 | 36 | 44 | 58
Not Completed | 4 | 6 | 3 | 2 | 6
Not completed — Adverse Event | 1 | 3 | 0 | 0 | 5
Not completed — Death | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 3 | 1 | 2 | 0
Not completed — Physician Decision | 2 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) | Arm B: Faricimab, 1.5 mg Q4W | Arm C: Faricimab, 6 mg Q4W | Arm D: Faricimab, 6 mg Every 4-8 Weeks | Arm E: Ranibizumab 0.5 mg + Faricimab 6 mg Q4W | Total
Number analyzed (Participants) | 68 | 46 | 39 | 46 | 64 | 263
Age, Continuous [Mean (Standard Deviation); unit: Years] | 76.4 (8.9) | 78.2 (8.9) | 78.0 (9.1) | 80.0 (8.0) | 79.2 (8.3) | 78.3 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 32 | 27 | 34 | 40 | 172
  Male | 29 | 14 | 12 | 12 | 24 | 91
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 0 | 4 | 2 | 13
  Not Hispanic or Latino | 64 | 43 | 38 | 42 | 61 | 248
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 0 | 1
  White | 66 | 45 | 39 | 44 | 64 | 258
  More than one race | 1 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 0 | 1 | 0 | 2
Best-Corrected Visual Acuity (BCVA) Letter Score in the Study Eye at Baseline [Mean (Standard Deviation); unit: BCVA Letters] — Best corrected visual acuity (BCVA) at a starting test distance of 4 meters was measured using a set of three Precision VisionTM or Lighthouse distance acuity charts (modified ETDRS Charts 1, 2, and R). The BCVA letter score for each participant ranges from 0 to 100 letters (best score attainable) correctly read on the acuity charts.
  BCVA Letters | 55.2 (12.7) | 56.7 (11.1) | 56.2 (12.2) | 56.3 (11.5) | 55.7 (11.6) | 55.9 (11.9)
Best-Corrected Visual Acuity (BCVA) Letter Score Category in the Study Eye at Baseline [Count of Participants; unit: Participants]
  BCVA Letter Score ≤54 | 22 | 20 | 15 | 21 | 26 | 104
  BCVA Letter Score >54 | 45 | 26 | 24 | 25 | 38 | 158
  Assessment Missing | 1 | 0 | 0 | 0 | 0 | 1
Choroidal Neovascularization (CNV) Lesion Type in the Study Eye at Baseline [Count of Participants; unit: Participants]
  Classic & Occult CNV | 26 | 19 | 12 | 20 | 21 | 98
  Classic CNV | 8 | 6 | 7 | 6 | 10 | 37
  Occult CNV | 33 | 20 | 20 | 19 | 33 | 125
  Assessment Missing | 1 | 1 | 0 | 1 | 0 | 3
Presence or Absence of Retinal Angiomatous Proliferation (RAP) in the Study Eye at Baseline [Count of Participants; unit: Participants]
  RAP Absent | 44 | 30 | 29 | 29 | 47 | 179
  RAP Present | 22 | 14 | 9 | 14 | 16 | 75
  Assessment Missing | 2 | 2 | 1 | 3 | 1 | 9
Presence or Absence of Polypoidal Choroidal Vasculopathy (PCV) in the Study Eye at Baseline [Count of Participants; unit: Participants]
  PCV Absent | 61 | 42 | 36 | 40 | 57 | 236
  PCV Present | 7 | 3 | 3 | 5 | 7 | 25
  Assessment Missing | 0 | 1 | 0 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in BCVA Letter Score at Week 36, in Treatment-Naive Participants
Description: Best corrected visual acuity (BCVA) at a starting test distance of 4 meters was measured using a set of three Precision VisionTM or Lighthouse distance acuity charts (modified ETDRS Charts 1, 2, and R) prior to dilating eyes by a trained and certified visual acuity examiner masked to study drug arm assignment. The BCVA examiner was masked to study eye and treatment assignment and only performed the refraction and BCVA assessment, but was not allowed to perform any other tasks involving direct care. The BCVA examiner was also masked to the BCVA letter scores of a participant's previous visits and could only know the refraction data from previous visits. The BCVA letter score ranges from 0 to 100 (best score attainable), and a gain in BCVA letter score from baseline indicates an improvement in visual acuity. The primary analysis used a Mixed Effects Model for Repeated Measurements (MMRM). Missing data were implicitly imputed by the MMRM, assuming a missing-at-random mechanism.
Time Frame: Baseline, Week 36
Population: Treatment-naive participants randomized to Arms A, B, C, and D.
Measure: Least Squares Mean (80% Confidence Interval); unit: BCVA Letters
Arm/Group | Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) | Arm B: Faricimab, 1.5 mg Q4W | Arm C: Faricimab, 6 mg Q4W | Arm D: Faricimab, 6 mg Every 4-8 Weeks
Number analyzed (Participants) | 68 | 46 | 39 | 46
BCVA Letters | 7.61 [5.43 to 9.80] | 9.18 [6.54 to 11.83] | 6.02 [3.24 to 8.80] | 6.10 [3.56 to 8.64]
Statistical Analysis 1: Comparison: Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) vs Arm B: Faricimab, 1.5 mg Q4W; The null hypothesis (Ho) was that there was no difference in means between the treatment group (Arm B) and the control group (Arm A). The alternative hypothesis (Ha) was that Arm B mean was different from Arm A mean; Test type: Superiority; p = 0.5244, Mixed Model for Repeated Measures — The threshold for statistical significance was an unadjusted 2-sided p-value <0.2. There was no formal correction for multiple comparisons; Categorical covariates(cov): RAP/PCV at baseline(BL), treatment group, visit, & visit by treatment group; Continuous cov: BCVA at BL; Unstructured cov; Difference in Least Squares Means = 1.57, 80% CI 2-sided [-1.60 to 4.74] — The mean difference was calculated as Arm B minus Arm A
Statistical Analysis 2: Comparison: Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) vs Arm C: Faricimab, 6 mg Q4W; The null hypothesis (Ho) was that there was no difference in means between the treatment group (Arm C) and the control group (Arm A). The alternative hypothesis (Ha) was that Arm C mean was different from Arm A mean; Test type: Superiority; p = 0.5308, Mixed Model for Repeated Measures — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = -1.59, 80% CI 2-sided [-4.86 to 1.67] — The mean difference was calculated as Arm C minus Arm A
Statistical Analysis 3: Comparison: Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) vs Arm D: Faricimab, 6 mg Every 4-8 Weeks; The null hypothesis (Ho) was that there was no difference in means between the treatment group (Arm D) and the control group (Arm A). The alternative hypothesis (Ha) was that Arm D mean was different from Arm A mean; Test type: Superiority; p = 0.5309, Mixed Model for Repeated Measures — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = -1.51, 80% CI 2-sided [-4.62 to 1.59] — The mean difference was calculated as Arm D minus Arm A

2. Primary Outcome: Mean Change From Week 12 in BCVA Letter Score at Week 36, in Anti-VEGF Incomplete Responders
Description: as for outcome 1
Time Frame: Weeks 12 and 36
Population: Anti-VEGF incomplete responders, which consisted of participants randomized to Arms A and E with BCVA ≤68 at Week 12 with at least one letter improvement relative to Baseline.
Measure: Least Squares Mean (80% Confidence Interval); unit: BCVA Letters
Arm/Group | Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) | Arm E: Ranibizumab 0.5 mg + Faricimab 6 mg Q4W
Number analyzed (Participants) | 37 | 38
BCVA Letters | 1.72 [-0.69 to 4.13] | 0.04 [-2.27 to 2.35]
Statistical Analysis 1: Comparison: Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) vs Arm E: Ranibizumab 0.5 mg + Faricimab 6 mg Q4W; The null hypothesis (Ho) was that there was no difference in means between the treatment group (Arm E) and the control group (Arm A). The alternative hypothesis (Ha) was that the Arm E mean was different from Arm A mean; Test type: Superiority; p = 0.3034, Mixed Model for Repeated Measures — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = -1.68, 80% CI 2-sided [-3.77 to 0.42] — The mean difference was calculated as Arm E minus Arm A

3. Secondary Outcome: Percentage of Participants Gaining Greater Than or Equal to (≥) 15 Letters From Baseline in BCVA Letter Score at Week 36, in Treatment-Naive Participants
Description: Best corrected visual acuity (BCVA) at a starting test distance of 4 meters was measured using a set of three Precision VisionTM or Lighthouse distance acuity charts (modified ETDRS Charts 1, 2, and R) prior to dilating eyes by a trained and certified visual acuity examiner masked to study drug arm assignment. The BCVA examiner was masked to study eye and treatment assignment and only performed the refraction and BCVA assessment, but was not allowed to perform any other tasks involving direct care. The BCVA examiner was also masked to the BCVA letter scores of a participant's previous visits and could only know the participant's refraction data from previous visits. The BCVA letter score ranges from 0 to 100 (best score attainable), and a gain in BCVA letter score from baseline indicates an improvement in visual acuity. The outcome measure was analyzed using a Generalized Estimating Equations Model. Missing values were not imputed; it was assumed that the data were missing at random.
Time Frame: Baseline, Week 36
Population: Treatment-naive participants randomized to Arms A, B, C, and D.
Measure: Least Squares Mean (80% Confidence Interval); unit: Percentage of Participants
Arm/Group | Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) | Arm B: Faricimab, 1.5 mg Q4W | Arm C: Faricimab, 6 mg Q4W | Arm D: Faricimab, 6 mg Every 4-8 Weeks
Number analyzed (Participants) | 68 | 46 | 39 | 46
Percentage of Participants | 31.0 [24.1 to 38.8] | 36.6 [27.6 to 46.7] | 27.9 [19.6 to 38.0] | 23.7 [16.5 to 32.7]
Statistical Analysis 1: Comparison: Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) vs Arm B: Faricimab, 1.5 mg Q4W; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.5527, Generalized Estimating Equations Model — [p-value comment as in outcome 1, analysis 1]; Categorical covariates: treatment group, visit, and visit by treatment group interaction. An AR(1) covariance structure was also used; Difference in Least Squares Means = 5.63, 80% CI 2-sided [-6.52 to 17.77] — The mean difference was calculated as Arm B minus Arm A
Statistical Analysis 2: Comparison: Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) vs Arm C: Faricimab, 6 mg Q4W; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.7382, Generalized Estimating Equations Model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 3, analysis 1]; Difference in Least Squares Means = -3.09, 80% CI 2-sided [-14.95 to 8.76] — The mean difference was calculated as Arm C minus Arm A
Statistical Analysis 3: Comparison: Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) vs Arm D: Faricimab, 6 mg Every 4-8 Weeks; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = 0.3932, Generalized Estimating Equations Model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 3, analysis 1]; Difference in Least Squares Means = -7.32, 80% CI 2-sided [-18.32 to 3.67] — The mean difference was calculated as Arm D minus Arm A

4. Secondary Outcome: Percentage of Participants Gaining ≥15 Letters From Week 12 in BCVA Letter Score at Week 36, in Anti-VEGF Incomplete Responders
Description: Best corrected visual acuity (BCVA) at a starting test distance of 4 meters was measured using a set of three Precision VisionTM or Lighthouse distance acuity charts (modified ETDRS Charts 1, 2, and R) prior to dilating eyes by a trained and certified visual acuity examiner masked to study drug arm assignment. The BCVA examiner was masked to study eye and treatment assignment and only performed the refraction and BCVA assessment, but was not allowed to perform any other tasks involving direct care. The BCVA examiner was also masked to the BCVA letter scores of a participant's previous visits and could only know the participant's refraction data from previous visits. The BCVA letter score ranges from 0 to 100 (best score attainable), and a gain in BCVA letter score from baseline indicates an improvement in visual acuity. Missing values were not imputed; it was assumed that the data were missing at random.
Time Frame: Weeks 12 and 36
Population: Anti-VEGF incomplete responders, which consisted of participants randomized to Arms A and E with BCVA ≤68 at Week 12 with at least one letter improvement relative to Baseline. This analysis only included participants with non-missing assessments at Weeks 12 and 36.
Measure: Number (80% Confidence Interval); unit: Percentage of Participants
Arm/Group | Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) | Arm E: Ranibizumab 0.5 mg + Faricimab 6 mg Q4W
Number analyzed (Participants) | 35 | 37
Percentage of Participants | 5.71 [0.69 to 10.74] | 0.00 [0.00 to 0.00]
Statistical Analysis 1: Comparison: Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) vs Arm E: Ranibizumab 0.5 mg + Faricimab 6 mg Q4W; The null hypothesis (Ho) was that there was no difference between the treatment group (Arm E) and the control group (Arm A). The alternative hypothesis (Ha) was that Arm E was different from Arm A; Test type: Superiority; p = 0.2328, Fisher Exact — [p-value comment as in outcome 1, analysis 1]; Difference in Percentage of Participants = -5.71, 80% CI 2-sided [-10.74 to -0.69] — The difference was calculated as Arm E minus Arm A

5. Secondary Outcome: Percentage of Participants With BCVA Snellen Equivalent of 20/40 or Better at Week 36, in Treatment-Naive Participants
Description: as for outcome 3
Time Frame: Week 36
Population: Treatment-naive participants randomized to Arms A, B, C, and D.
Measure: Least Squares Mean (80% Confidence Interval); unit: Percentage of Participants
Arm/Group | Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) | Arm B: Faricimab, 1.5 mg Q4W | Arm C: Faricimab, 6 mg Q4W | Arm D: Faricimab, 6 mg Every 4-8 Weeks
Number analyzed (Participants) | 68 | 46 | 39 | 46
Percentage of Participants | 49.5 [41.6 to 57.4] | 49.0 [39.2 to 58.8] | 39.4 [29.8 to 49.9] | 41.8 [32.8 to 51.4]
Statistical Analysis 1: Comparison: Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) vs Arm B: Faricimab, 1.5 mg Q4W; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.9581, Generalized Estimating Equations Model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 3, analysis 1]; Difference in Least Squares Means = -0.52, 80% CI 2-sided [-13.26 to 12.22] — The mean difference was calculated as Arm B minus Arm A
Statistical Analysis 2: Comparison: Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) vs Arm C: Faricimab, 6 mg Q4W; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.3166, Generalized Estimating Equations Model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 3, analysis 1]; Difference in Least Squares Means = -10.08, 80% CI 2-sided [-22.99 to 2.82] — The mean difference was calculated as Arm C minus Arm A
Statistical Analysis 3: Comparison: Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) vs Arm D: Faricimab, 6 mg Every 4-8 Weeks; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = 0.4244, Generalized Estimating Equations Model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 3, analysis 1]; Difference in Least Squares Means = -7.68, 80% CI 2-sided [-20.01 to 4.64] — The mean difference was calculated as Arm D minus Arm A

6. Secondary Outcome: Percentage of Participants With BCVA Snellen Equivalent of 20/40 or Better at Week 36, in Anti-VEGF Incomplete Responders
Description: as for outcome 4
Time Frame: Week 36
Population: Anti-VEGF incomplete responders, which consisted of participants randomized to Arms A and E with BCVA ≤68 at Week 12 with at least one letter improvement relative to Baseline. This analysis only included participants with non-missing assessments at Week 36.
Measure: Number (80% Confidence Interval); unit: Percentage of Participants
Arm/Group | Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) | Arm E: Ranibizumab 0.5 mg + Faricimab 6 mg Q4W
Number analyzed (Participants) | 35 | 37
Percentage of Participants | 22.86 [13.76 to 31.95] | 16.22 [8.45 to 23.98]
Statistical Analysis 1: Comparison: Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) vs Arm E: Ranibizumab 0.5 mg + Faricimab 6 mg Q4W; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.5586, Fisher Exact — [p-value comment as in outcome 1, analysis 1]; Difference in Percentage of Participants = -6.64, 80% CI 2-sided [-18.60 to 5.32] — The difference was calculated as Arm E minus Arm A

7. Secondary Outcome: Percentage of Participants With BCVA Snellen Equivalent of 20/200 or Worse at Week 36, in Treatment-Naive Participants
Description: as for outcome 3
Time Frame: Week 36
Population: Treatment-naive participants randomized to Arms A, B, C, and D.
Measure: Least Squares Mean (80% Confidence Interval); unit: Percentage of Participants
Arm/Group | Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) | Arm B: Faricimab, 1.5 mg Q4W | Arm C: Faricimab, 6 mg Q4W | Arm D: Faricimab, 6 mg Every 4-8 Weeks
Number analyzed (Participants) | 68 | 46 | 39 | 46
Percentage of Participants | 7.7 [4.4 to 13.2] | 8.7 [4.6 to 16.0] | 15.8 [9.6 to 25.0] | 8.8 [4.7 to 15.9]
Statistical Analysis 1: Comparison: Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) vs Arm B: Faricimab, 1.5 mg Q4W; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.8536, Generalized Estimating Equations Model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 3, analysis 1]; Difference in Least Squares Means = 1.00, 80% CI 2-sided [-5.93 to 7.93] — The mean difference was calculated as Arm B minus Arm A
Statistical Analysis 2: Comparison: Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) vs Arm C: Faricimab, 6 mg Q4W; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.2303, Generalized Estimating Equations Model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 3, analysis 1]; Difference in Least Squares Means = 8.14, 80% CI 2-sided [-0.56 to 16.83] — The mean difference was calculated as Arm C minus Arm A
Statistical Analysis 3: Comparison: Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) vs Arm D: Faricimab, 6 mg Every 4-8 Weeks; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = 0.8406, Generalized Estimating Equations Model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 3, analysis 1]; Difference in Least Squares Means = 1.08, 80% CI 2-sided [-5.79 to 7.95] — The mean difference was calculated as Arm D minus Arm A

8. Secondary Outcome: Percentage of Participants With BCVA Snellen Equivalent of 20/200 or Worse at Week 36, in Anti-VEGF Incomplete Responders
Description: as for outcome 4
Time Frame: Week 36
Population: as for outcome 6
Measure: Number (80% Confidence Interval); unit: Percentage of Participants
Arm/Group | Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) | Arm E: Ranibizumab 0.5 mg + Faricimab 6 mg Q4W
Number analyzed (Participants) | 35 | 37
Percentage of Participants | 14.29 [6.71 to 21.87] | 13.51 [6.31 to 20.72]
Statistical Analysis 1: Comparison: Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) vs Arm E: Ranibizumab 0.5 mg + Faricimab 6 mg Q4W; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 1.0000, Fisher Exact — [p-value comment as in outcome 1, analysis 1]; Difference in Percentage of Participants = -0.77, 80% CI 2-sided [-11.23 to 9.68] — The difference was calculated as Arm E minus Arm A

9. Secondary Outcome: Mean Change From Baseline in Foveal Center Point Thickness at Week 36, as Measured by Spectral Domain Optical Coherence Tomography (SD-OCT), in Treatment-Naive Participants
Description: Foveal center point thickness (FCPT) is defined as the thickness from the inner limiting membrane to the retinal pigment epithelial at the horizontal slice closest to the center of the fovea. Foveal center point thickness was measured using spectral domain optical coherence tomography (SD-OCT). Anatomic outcome measures were based on results from a central reading center. This analysis used a Mixed Effects Model for Repeated Measurements (MMRM). Missing data were implicitly imputed by the MMRM, assuming a missing-at-random mechanism.
Time Frame: Baseline, Week 36
Population: Treatment-naive participants randomized to Arms A, B, C, and D.
Measure: Least Squares Mean (80% Confidence Interval); unit: micrometres (μm)
Arm/Group | Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) | Arm B: Faricimab, 1.5 mg Q4W | Arm C: Faricimab, 6 mg Q4W | Arm D: Faricimab, 6 mg Every 4-8 Weeks
Number analyzed (Participants) | 68 | 46 | 39 | 46
micrometres (μm) | -194.00 [-207.01 to -181.00] | -181.35 [-196.90 to -165.81] | -193.12 [-209.49 to -176.76] | -161.20 [-176.15 to -146.25]
Statistical Analysis 1: Comparison: Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) vs Arm B: Faricimab, 1.5 mg Q4W; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.3798, Mixed Model for Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Categorical covariates(cov): RAP/PCV at baseline(BL), treatment group, visit, & visit by treatment group; Continuous cov: FCPT at BL; Unstructured cov; Difference in Least Squares Means = 12.65, 80% CI 2-sided [-5.81 to 31.11] — The mean difference was calculated as Arm B minus Arm A
Statistical Analysis 2: Comparison: Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) vs Arm C: Faricimab, 6 mg Q4W; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.9529, Mixed Model for Repeated Measures — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 9, analysis 1]; Difference in Least Squares Means = 0.88, 80% CI 2-sided [-18.3 to 20.03] — The mean difference was calculated as Arm C minus Arm A
Statistical Analysis 3: Comparison: Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) vs Arm D: Faricimab, 6 mg Every 4-8 Weeks; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = 0.0208, Mixed Model for Repeated Measures — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 9, analysis 1]; Difference in Least Squares Means = 32.81, 80% CI 2-sided [14.65 to 50.96] — The mean difference was calculated as Arm D minus Arm A

10. Secondary Outcome: Mean Change From Week 12 in Foveal Center Point Thickness at Week 36, as Measured by SD-OCT, in Anti-VEGF Incomplete Responders
Description: as for outcome 9
Time Frame: Weeks 12 and 36
Population: as for outcome 2
Measure: Least Squares Mean (80% Confidence Interval); unit: micrometres (μm)
Arm/Group | Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) | Arm E: Ranibizumab 0.5 mg + Faricimab 6 mg Q4W
Number analyzed (Participants) | 37 | 38
micrometres (μm) | -14.5 [-28.7 to -0.2] | -20.8 [-34.5 to -7.1]
Statistical Analysis 1: Comparison: Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) vs Arm E: Ranibizumab 0.5 mg + Faricimab 6 mg Q4W; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.5185, Mixed Model for Repeated Measures — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 9, analysis 1]; Difference in Least Squares Means = -6.35, 80% CI 2-sided [-19.0 to 6.27] — The mean difference was calculated as Arm E minus Arm A

11. Secondary Outcome: Mean Change From Baseline in Central Subfield Thickness at Week 36, as Measured by SD-OCT, in Treatment-Naive Participants
Description: Central subfield thickness (CST) is defined as the mean thickness from the inner limiting membrane to the retinal pigment epithelial over the 1 millimetre (mm) central subfield. Central subfield thickness was measured using spectral domain optical coherence tomography (SD-OCT). Anatomic outcome measures were based on results from a central reading center. This analysis used a Mixed Effects Model for Repeated Measurements (MMRM). Missing data were implicitly imputed by the MMRM, assuming a missing-at-random mechanism.
Time Frame: Baseline, Week 36
Population: Treatment-naive participants randomized to Arms A, B, C, and D.
Measure: Least Squares Mean (80% Confidence Interval); unit: micrometres (μm)
Arm/Group | Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) | Arm B: Faricimab, 1.5 mg Q4W | Arm C: Faricimab, 6 mg Q4W | Arm D: Faricimab, 6 mg Every 4-8 Weeks
Number analyzed (Participants) | 68 | 46 | 39 | 46
micrometres (μm) | -176.18 [-188.94 to -163.43] | -156.73 [-171.85 to -141.61] | -173.40 [-189.40 to -157.40] | -147.66 [-162.27 to -133.05]
Statistical Analysis 1: Comparison: Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) vs Arm B: Faricimab, 1.5 mg Q4W; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.1624, Mixed Model for Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Categorical covariates(cov): RAP/PCV at baseline(BL), treatment group, visit, & visit by treatment group; Continuous cov: CST at BL; Unstructured cov; Difference in Least Squares Means = 19.45, 80% CI 2-sided [1.61 to 37.29] — The mean difference was calculated as Arm B minus Arm A
Statistical Analysis 2: Comparison: Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) vs Arm C: Faricimab, 6 mg Q4W; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.8475, Mixed Model for Repeated Measures — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 11, analysis 1]; Difference in Least Squares Means = 2.79, 80% CI 2-sided [-15.8 to 21.37] — The mean difference was calculated as Arm C minus Arm A
Statistical Analysis 3: Comparison: Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) vs Arm D: Faricimab, 6 mg Every 4-8 Weeks; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = 0.0381, Mixed Model for Repeated Measures — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 11, analysis 1]; Difference in Least Squares Means = 28.52, 80% CI 2-sided [10.93 to 46.11] — The mean difference was calculated as Arm D minus Arm A

12. Secondary Outcome: Mean Change From Week 12 in Central Subfield Thickness at Week 36, as Measured by SD-OCT in Anti-VEGF Incomplete Responders
Description: as for outcome 11
Time Frame: Weeks 12 and 36
Population: as for outcome 2
Measure: Least Squares Mean (80% Confidence Interval); unit: micrometres (μm)
Arm/Group | Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) | Arm E: Ranibizumab 0.5 mg + Faricimab 6 mg Q4W
Number analyzed (Participants) | 37 | 38
micrometres (μm) | -17.00 [-33.12 to -0.88] | -31.42 [-46.83 to -16.02]
Statistical Analysis 1: Comparison: Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) vs Arm E: Ranibizumab 0.5 mg + Faricimab 6 mg Q4W; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.2089, Mixed Model for Repeated Measures — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 11, analysis 1]; Difference in Least Squares Means = -14.4, 80% CI 2-sided [-29.1 to 0.29] — The mean difference was calculated as Arm E minus Arm A

13. Secondary Outcome: Number of Participants With Resolution of Dry Retina at Week 36, Defined as Absence of Cysts, Intraretinal Fluid, Pigment Epithelial Detachment, or Subretinal Fluid as Measured by SD-OCT, in Treatment-Naive Participants
Description: The presence of cysts, intraretinal fluid, pigment epithelial detachment, or subretinal fluid, as per the study's dry retina definition, were evaluated as individual dry retina outcomes. Cysts were defined as the presence of cystoid space (fluid) in the retina. Intraretinal fluid was defined as the presence of fluid within the retina. Pigment epithelial detachment was defined as the presence of a detachment of the pigment epithelium from the Bruch's membrane. Subretinal fluid was defined as the presence of fluid between the retina and the retinal pigment epithelium. All parameters were measured using spectral domain optical coherence tomography (SD-OCT). Anatomic outcome measures were based on results from a central reading center.
Time Frame: Baseline, Week 36
Population: Treatment-naive participants randomized to Arms A, B, C, and D. This analysis only included participants with presence of the individual dry retina measures (cysts, intraretinal fluid, pigment epithelial detachment, or subretinal fluid) at Baseline and who were reassessed at Week 36.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) | Arm B: Faricimab, 1.5 mg Q4W | Arm C: Faricimab, 6 mg Q4W | Arm D: Faricimab, 6 mg Every 4-8 Weeks
Number analyzed (Participants) | 68 | 46 | 39 | 46
Participants
  Cysts: Present at Baseline: number analyzed (Participants) | 52 | 29 | 29 | 38
  Cysts: Present at Baseline | 52 | 29 | 29 | 38
  Cysts: Present at Week 36: number analyzed (Participants) | 49 | 25 | 27 | 36
  Cysts: Present at Week 36 | 13 | 7 | 6 | 11
  Cysts: Absent at Week 36: number analyzed (Participants) | 49 | 25 | 27 | 36
  Cysts: Absent at Week 36 | 36 | 18 | 21 | 25
  Intraretinal Fluid: Present at Baseline: number analyzed (Participants) | 67 | 46 | 39 | 45
  Intraretinal Fluid: Present at Baseline | 67 | 46 | 39 | 45
  Intraretinal Fluid: Present at Week 36: number analyzed (Participants) | 64 | 40 | 37 | 43
  Intraretinal Fluid: Present at Week 36 | 46 | 27 | 28 | 34
  Intraretinal Fluid: Absent at Week 36: number analyzed (Participants) | 64 | 40 | 39 | 46
  Intraretinal Fluid: Absent at Week 36 | 18 | 13 | 9 | 9
  Pigment Epithelial Detachment: Present at Baseline: number analyzed (Participants) | 58 | 37 | 27 | 36
  Pigment Epithelial Detachment: Present at Baseline | 58 | 37 | 27 | 36
  Pigment Epithelial Detachment: Present at Week 36: number analyzed (Participants) | 55 | 31 | 26 | 36
  Pigment Epithelial Detachment: Present at Week 36 | 43 | 25 | 20 | 32
  Pigment Epithelial Detachment: Absent at Week 36: number analyzed (Participants) | 55 | 31 | 26 | 36
  Pigment Epithelial Detachment: Absent at Week 36 | 12 | 6 | 6 | 4
  Subretinal Fluid: Present at Baseline: number analyzed (Participants) | 56 | 41 | 30 | 35
  Subretinal Fluid: Present at Baseline | 56 | 41 | 30 | 35
  Subretinal Fluid: Present at Week 36: number analyzed (Participants) | 53 | 36 | 29 | 33
  Subretinal Fluid: Present at Week 36 | 11 | 18 | 3 | 8
  Subretinal Fluid: Absent at Week 36: number analyzed (Participants) | 53 | 36 | 29 | 33
  Subretinal Fluid: Absent at Week 36 | 42 | 18 | 26 | 25

14. Secondary Outcome: Number of Participants With Resolution of Dry Retina at Week 36, Defined as Absence of Cysts, Intraretinal Fluid, Pigment Epithelial Detachment, or Subretinal Fluid as Measured by SD-OCT, in Anti-VEGF Incomplete Responders
Description: as for outcome 13
Time Frame: Weeks 12 and 36
Population: Anti-VEGF incomplete responders, consisting of participants randomized to Arms A and E with BCVA ≤68 at Week 12 with ≥1 letter increase from Baseline. Analysis only included those with presence of individual dry retina measures (cysts, intraretinal fluid, pigment epithelial detachment, or subretinal fluid) at Week 12 and reassessed at Week 36.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) | Arm E: Ranibizumab 0.5 mg + Faricimab 6 mg Q4W
Number analyzed (Participants) | 37 | 38
Participants
  Cysts: Present at Week 12: number analyzed (Participants) | 9 | 11
  Cysts: Present at Week 12 | 9 | 11
  Cysts: Present at Week 36: number analyzed (Participants) | 9 | 11
  Cysts: Present at Week 36 | 4 | 5
  Cysts: Absent at Week 36: number analyzed (Participants) | 9 | 11
  Cysts: Absent at Week 36 | 5 | 6
  Intraretinal Fluid: Present at Week 12: number analyzed (Participants) | 28 | 36
  Intraretinal Fluid: Present at Week 12 | 28 | 36
  Intraretinal Fluid: Present at Week 36: number analyzed (Participants) | 26 | 35
  Intraretinal Fluid: Present at Week 36 | 19 | 28
  Intraretinal Fluid: Absent at Week 36: number analyzed (Participants) | 26 | 35
  Intraretinal Fluid: Absent at Week 36 | 7 | 7
  Pigment Epithelial Detachment: Present at Week 12: number analyzed (Participants) | 24 | 28
  Pigment Epithelial Detachment: Present at Week 12 | 24 | 28
  Pigment Epithelial Detachment: Present at Week 36: number analyzed (Participants) | 22 | 27
  Pigment Epithelial Detachment: Present at Week 36 | 19 | 22
  Pigment Epithelial Detachment: Absent at Week 36: number analyzed (Participants) | 22 | 27
  Pigment Epithelial Detachment: Absent at Week 36 | 3 | 5
  Subretinal Fluid: Present at Week 12: number analyzed (Participants) | 10 | 9
  Subretinal Fluid: Present at Week 12 | 10 | 9
  Subretinal Fluid: Present at Week 36: number analyzed (Participants) | 8 | 8
  Subretinal Fluid: Present at Week 36 | 3 | 2
  Subretinal Fluid: Absent at Week 36: number analyzed (Participants) | 8 | 8
  Subretinal Fluid: Absent at Week 36 | 5 | 6

15. Secondary Outcome: Mean Change From Baseline in Total Area of Choroidal Neovascularization (CNV) at Week 36, as Measured by Fundus Fluorescein Angiography (FFA), in Treatment-Naive Participants
Description: The total area of choroidal neovascularization (CNV) was evaluated by a central reading center using fundus fluorescein angiography (FFA). This analysis used a Mixed Effects Model for Repeated Measurements (MMRM). Missing data were implicitly imputed by the MMRM, assuming a missing-at-random mechanism.
Time Frame: Baseline, Week 36
Population: Treatment-naive participants randomized to Arms A, B, C, and D.
Measure: Least Squares Mean (80% Confidence Interval); unit: millimetres squared (mm^2)
Arm/Group | Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) | Arm B: Faricimab, 1.5 mg Q4W | Arm C: Faricimab, 6 mg Q4W | Arm D: Faricimab, 6 mg Every 4-8 Weeks
Number analyzed (Participants) | 68 | 46 | 39 | 46
millimetres squared (mm^2) | -3.41 [-4.34 to -2.49] | -3.81 [-4.93 to -2.70] | -3.19 [-4.29 to -2.08] | -3.31 [-4.31 to -2.30]
Statistical Analysis 1: Comparison: Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) vs Arm B: Faricimab, 1.5 mg Q4W; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.6717, Mixed Model for Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Categorical covariates(cov): RAP/PCV at baseline(BL), treatment group, visit, & visit by treatment group; Continuous cov: CNV at BL; Unstructured cov; Difference in Least Squares Means = -0.40, 80% CI 2-sided [-1.61 to 0.81] — The mean difference was calculated as Arm B minus Arm A
Statistical Analysis 2: Comparison: Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) vs Arm C: Faricimab, 6 mg Q4W; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.8131, Mixed Model for Repeated Measures — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 15, analysis 1]; Difference in Least Squares Means = 0.23, 80% CI 2-sided [-1.01 to 1.47] — The mean difference was calculated as Arm C minus Arm A
Statistical Analysis 3: Comparison: Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) vs Arm D: Faricimab, 6 mg Every 4-8 Weeks; The null hypothesis (Ho) was that there was no difference in means between each of the treatment groups (Arms B, C, or D) and the control group (Arm A). The alternative hypothesis (Ha) was that Arms B, C, or D means were different from Arm A mean; Test type: Superiority; p = 0.9069, Mixed Model for Repeated Measures — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 15, analysis 1]; Difference in Least Squares Means = 0.11, 80% CI 2-sided [-1.07 to 1.29] — The mean difference was calculated as Arm D minus Arm A

16. Secondary Outcome: Mean Change From Week 12 in Total Area of Choroidal Neovascularization (CNV) at Week 36, as Measured by FFA, in Anti-VEGF Incomplete Responders
Description: The total area of choroidal neovascularization (CNV) was evaluated by a central reading center using fundus fluorescein angiography (FFA).
Time Frame: Weeks 12 and 36
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: millimetres squared (mm^2)
Arm/Group | Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) | Arm E: Ranibizumab 0.5 mg + Faricimab 6 mg Q4W
Number analyzed (Participants) | 22 | 21
millimetres squared (mm^2) | -0.50 (2.37) | -1.37 (3.72)

17. Secondary Outcome: Mean Change From Baseline in Total Area of Choroidal Neovascularization (CNV) Component at Week 36, as Measured by FFA, in Treatment-Naive Participants
Description: The total area of choroidal neovascularization (CNV) component (i.e., total area of CNV membrane) was evaluated by a central reading center using fundus fluorescein angiography (FFA). This analysis used a Mixed Effects Model for Repeated Measurements (MMRM). Missing data were implicitly imputed by the MMRM, assuming a missing-at-random mechanism.
Time Frame: Baseline, Week 36
Population: Treatment-naive participants randomized to Arms A, B, C, and D.
Measure: Least Squares Mean (80% Confidence Interval); unit: millimetres squared (mm^2)
Arm/Group | Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) | Arm B: Faricimab, 1.5 mg Q4W | Arm C: Faricimab, 6 mg Q4W | Arm D: Faricimab, 6 mg Every 4-8 Weeks
Number analyzed (Participants) | 68 | 46 | 39 | 46
millimetres squared (mm^2) | -4.18 [-5.09 to -3.27] | -5.14 [-6.24 to -4.04] | -2.96 [-4.09 to -1.82] | -3.83 [-4.84 to -2.82]
Statistical Analysis 1: Comparison: Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) vs Arm B: Faricimab, 1.5 mg Q4W; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.3189, Mixed Model for Repeated Measures — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 15, analysis 1]; Difference in Least Squares Means = -0.96, 80% CI 2-sided [-2.20 to 0.28] — The mean difference was calculated as Arm B minus Arm A
Statistical Analysis 2: Comparison: Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) vs Arm C: Faricimab, 6 mg Q4W; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.2256, Mixed Model for Repeated Measures — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 15, analysis 1]; Difference in Least Squares Means = 1.22, 80% CI 2-sided [-0.07 to 2.52] — The mean difference was calculated as Arm C minus Arm A
Statistical Analysis 3: Comparison: Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) vs Arm D: Faricimab, 6 mg Every 4-8 Weeks; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = 0.7086, Mixed Model for Repeated Measures — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 15, analysis 1]; Difference in Least Squares Means = 0.35, 80% CI 2-sided [-0.86 to 1.57] — The mean difference was calculated as Arm D minus Arm A

18. Secondary Outcome: Mean Change From Week 12 in Total Area of Choroidal Neovascularization (CNV) Component at Week 36, as Measured by FFA, in Anti-VEGF Incomplete Responders
Description: The total area of choroidal neovascularization (CNV) component (i.e., total area of CNV membrane) was evaluated by a central reading center using fundus fluorescein angiography (FFA).
Time Frame: Weeks 12 and 36
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: millimetres squared (mm^2)
Arm/Group | Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) | Arm E: Ranibizumab 0.5 mg + Faricimab 6 mg Q4W
Number analyzed (Participants) | 22 | 21
millimetres squared (mm^2) | -1.87 (4.05) | -1.88 (3.98)

19. Secondary Outcome: Mean Change From Baseline in Total Area of Leakage at Week 36, as Measured by FFA, in Treatment-Naive Participants
Description: The total area of leakage was evaluated by a central reading center using fundus fluorescein angiography (FFA). This analysis used a Mixed Effects Model for Repeated Measurements (MMRM). Missing data were implicitly imputed by the MMRM, assuming a missing-at-random mechanism.
Time Frame: Baseline, Week 36
Population: Treatment-naive participants randomized to Arms A, B, C, and D.
Measure: Least Squares Mean (80% Confidence Interval); unit: millimetres squared (mm^2)
Arm/Group | Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) | Arm B: Faricimab, 1.5 mg Q4W | Arm C: Faricimab, 6 mg Q4W | Arm D: Faricimab, 6 mg Every 4-8 Weeks
Number analyzed (Participants) | 68 | 46 | 39 | 46
millimetres squared (mm^2) | -5.15 [-6.10 to -4.20] | -5.94 [-7.10 to -4.77] | -3.71 [-4.88 to -2.53] | -4.66 [-5.70 to -3.61]
Statistical Analysis 1: Comparison: Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) vs Arm B: Faricimab, 1.5 mg Q4W; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.4353, Mixed Model for Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Categorical covariates(cov): RAP/PCV at baseline(BL), treatment group, visit, & visit by treatment group; Continuous cov: leak at BL; Unstructured cov; Difference in Least Squares Means = -0.78, 80% CI 2-sided [-2.07 to 0.51] — The mean difference was calculated as Arm B minus Arm A
Statistical Analysis 2: Comparison: Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) vs Arm C: Faricimab, 6 mg Q4W; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.1652, Mixed Model for Repeated Measures — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 19, analysis 1]; Difference in Least Squares Means = 1.45, 80% CI 2-sided [0.11 to 2.78] — The mean difference was calculated as Arm C minus Arm A
Statistical Analysis 3: Comparison: Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) vs Arm D: Faricimab, 6 mg Every 4-8 Weeks; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = 0.61111, Mixed Model for Repeated Measures — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 19, analysis 1]; Difference in Least Squares Means = 0.50, 80% CI 2-sided [-0.76 to 1.75] — The mean difference was calculated as Arm D minus Arm A

20. Secondary Outcome: Mean Change From Week 12 in Total Area of Leakage at Week 36, as Measured by FFA, in Anti-VEGF Incomplete Responders
Description: The total area of leakage was evaluated by a central reading center using fundus fluorescein angiography (FFA).
Time Frame: Weeks 12 and 36
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: millimetres squared (mm^2)
Arm/Group | Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) | Arm E: Ranibizumab 0.5 mg + Faricimab 6 mg Q4W
Number analyzed (Participants) | 22 | 21
millimetres squared (mm^2) | -1.87 (4.05) | -2.00 (3.98)

21. Secondary Outcome: Safety Summary of the Overall Number of Participants With at Least One Adverse Event by Event Type, in All Participants
Description: This safety summary reports the number and percentage of participants who experienced at least one adverse event (AE) during the study. AEs are categorized as any AEs, ocular AEs occurring in the study eye or fellow eye, systemic AEs, serious AEs, AEs related to treatment with study drug, AEs leading to discontinuation (withdrawal) of treatment with study drug, and AEs with fatal outcome. The investigator independently assessed the seriousness and severity for each AE. Severity was graded according to the following grading scale: Mild = Discomfort noticed, but no disruption of normal daily activity; Moderate = Discomfort sufficient to reduce or affect normal daily activity; Severe = Incapacitating with inability to work or to perform normal daily activity. Severity and seriousness are not synonymous; regardless of severity, some AEs may have also met seriousness criteria.
Time Frame: From Baseline until 28 days after the last dose of study treatment (up to 36 weeks)
Population: Safety Population: all participants who received at least one dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) | Arm B: Faricimab, 1.5 mg Q4W | Arm C: Faricimab, 6 mg Q4W | Arm D: Faricimab, 6 mg Every 4-8 Weeks | Arm E: Ranibizumab 0.5 mg + Faricimab 6 mg Q4W
Number analyzed (Participants) | 67 | 46 | 39 | 46 | 64
Participants
  Any Adverse Event (AE) | 51 | 39 | 31 | 39 | 54
  Ocular AE in Either Eye | 39 | 25 | 23 | 29 | 37
  Ocular AE in the Study Eye | 28 | 21 | 21 | 27 | 28
  Ocular AE in the Fellow Eye | 21 | 16 | 9 | 18 | 20
  Serious Ocular AE in the Study Eye | 0 | 3 | 0 | 0 | 2
  Ocular AE in Study Eye Leading to Withdrawal | 0 | 1 | 0 | 0 | 4
  Systemic AE | 37 | 37 | 23 | 30 | 43
  Serious Systemic AE | 9 | 7 | 7 | 4 | 6
  Systemic AE Leading to Withdrawal | 1 | 2 | 0 | 0 | 2
  AE with Fatal Outcome | 0 | 0 | 0 | 0 | 1
  Any Serious AE | 9 | 11 | 7 | 5 | 8
  Any Related Serious AE | 0 | 1 | 0 | 0 | 0
  Any Related AE | 3 | 4 | 3 | 3 | 0
  Related Ocular AE in the Study Eye | 3 | 4 | 3 | 3 | 0
  Related Systemic AE | 0 | 0 | 0 | 0 | 0

22. Secondary Outcome: Number of Participants With at Least One Ocular Adverse Event in the Study Eye or the Fellow Eye by Highest Intensity, in All Participants
Description: The investigator assessed adverse event severity according to the following grading scale: Mild = Discomfort noticed, but no disruption of normal daily activity; Moderate = Discomfort sufficient to reduce or affect normal daily activity; Severe = Incapacitating with inability to work or to perform normal daily activity. Only the most severe intensity was counted for multiple occurrences of the same adverse event per participant at the preferred term level. Severity and seriousness are not synonymous; regardless of severity, some adverse events may have also met seriousness criteria.
Time Frame: From Baseline until 28 days after the last dose of study treatment (up to 36 weeks)
Population: Safety Population: all participants who received at least one dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) | Arm B: Faricimab, 1.5 mg Q4W | Arm C: Faricimab, 6 mg Q4W | Arm D: Faricimab, 6 mg Every 4-8 Weeks | Arm E: Ranibizumab 0.5 mg + Faricimab 6 mg Q4W
Number analyzed (Participants) | 67 | 46 | 39 | 46 | 64
Participants
  Study Eye - Adverse Event (AE) of Any Grade | 28 | 21 | 21 | 27 | 28
  Study Eye - Mild AE | 27 | 19 | 20 | 25 | 24
  Study Eye - Moderate AE | 4 | 2 | 3 | 6 | 8
  Study Eye - Severe AE | 0 | 3 | 0 | 0 | 2
  Fellow Eye - AE of Any Grade | 21 | 16 | 9 | 18 | 20
  Fellow Eye - Mild AE | 15 | 14 | 7 | 17 | 17
  Fellow Eye - Moderate AE | 5 | 1 | 4 | 1 | 2
  Fellow Eye - Severe AE | 1 | 1 | 0 | 0 | 2

23. Secondary Outcome: Number of Participants With at Least One Systemic Adverse Event by Highest Intensity, in All Participants
Description: as for outcome 22
Time Frame: From Baseline until 28 days after the last dose of study treatment (up to 36 weeks)
Population: Safety Population: all participants who received at least one dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) | Arm B: Faricimab, 1.5 mg Q4W | Arm C: Faricimab, 6 mg Q4W | Arm D: Faricimab, 6 mg Every 4-8 Weeks | Arm E: Ranibizumab 0.5 mg + Faricimab 6 mg Q4W
Number analyzed (Participants) | 67 | 46 | 39 | 46 | 64
Participants
  Any Grade | 37 | 37 | 23 | 30 | 43
  Mild | 30 | 27 | 17 | 23 | 28
  Moderate | 16 | 18 | 14 | 13 | 26
  Severe | 7 | 2 | 5 | 4 | 4

24. Secondary Outcome: Number of Participants With Abnormal Systolic Blood Pressure, in All Participants
Description: Abnormal systolic blood pressure (supine) was defined as any value outside of the standard reference range, from <70 (low) to >140 (high) millimetres of mercury (mmHg). Baseline was defined as the last non-missing predose assessment. Not every abnormal vital sign qualified as an adverse event, only if it met any of the following criteria: clinically significant (per investigator); accompanied by clinical symptoms; resulted in a change in study treatment; or required a change in concomitant therapy.
Time Frame: Assessed at each study visit from Baseline until 28 days after the last dose of study treatment (up to 36 weeks)
Population: Safety Population: all participants who received at least one dose of study treatment. In this analysis, the number of participants with an abnormal vital sign (numerator) is reported among the number analyzed (denominator), which represents the number of participants without the abnormal vital sign at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) | Arm B: Faricimab, 1.5 mg Q4W | Arm C: Faricimab, 6 mg Q4W | Arm D: Faricimab, 6 mg Every 4-8 Weeks | Arm E: Ranibizumab 0.5 mg + Faricimab 6 mg Q4W
Number analyzed (Participants) | 67 | 46 | 39 | 46 | 64
Participants
  Low | 0 | 0 | 0 | 0 | 0
  High: number analyzed (Participants) | 43 | 24 | 22 | 29 | 37
  High | 20 | 13 | 13 | 23 | 25

25. Secondary Outcome: Number of Participants With Abnormal Diastolic Blood Pressure, in All Participants
Description: Abnormal diastolic blood pressure (supine) was defined as any value outside of the standard reference range, from <40 (low) to >90 (high) millimetres of mercury (mmHg). Baseline was defined as the last non-missing predose assessment. Not every abnormal vital sign qualified as an adverse event, only if it met any of the following criteria: clinically significant (per investigator); accompanied by clinical symptoms; resulted in a change in study treatment; or required a change in concomitant therapy.
Time Frame: Assessed at each study visit from Baseline until 28 days after the last dose of study treatment (up to 36 weeks)
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) | Arm B: Faricimab, 1.5 mg Q4W | Arm C: Faricimab, 6 mg Q4W | Arm D: Faricimab, 6 mg Every 4-8 Weeks | Arm E: Ranibizumab 0.5 mg + Faricimab 6 mg Q4W
Number analyzed (Participants) | 67 | 46 | 39 | 46 | 64
Participants
  Low | 0 | 0 | 0 | 0 | 0
  High: number analyzed (Participants) | 62 | 41 | 35 | 44 | 57
  High | 15 | 9 | 8 | 10 | 9

26. Secondary Outcome: Number of Participants With Abnormal Heart Rate, in All Participants
Description: Abnormal heart rate (supine) was defined as any value outside of the standard reference range, from <40 (low) to >100 (high) beats per minute. Baseline was defined as the last non-missing predose assessment. Not every abnormal vital sign qualified as an adverse event, only if it met any of the following criteria: clinically significant (per investigator); accompanied by clinical symptoms; resulted in a change in study treatment; or required a change in concomitant therapy.
Time Frame: Assessed at each study visit from Baseline until 28 days after the last dose of study treatment (up to 36 weeks)
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) | Arm B: Faricimab, 1.5 mg Q4W | Arm C: Faricimab, 6 mg Q4W | Arm D: Faricimab, 6 mg Every 4-8 Weeks | Arm E: Ranibizumab 0.5 mg + Faricimab 6 mg Q4W
Number analyzed (Participants) | 67 | 46 | 39 | 46 | 64
Participants
  Low | 1 | 0 | 1 | 0 | 0
  High: number analyzed (Participants) | 65 | 46 | 39 | 46 | 63
  High | 1 | 0 | 1 | 1 | 1

27. Secondary Outcome: Number of Participants With Abnormal Body Temperature, in All Participants
Description: Abnormal body temperature (supine) was defined as any value outside of the standard reference range, from <36.5 (low) to >37.5 (high) degrees Celsius. Baseline was defined as the last non-missing predose assessment. Not every abnormal vital sign qualified as an adverse event, only if it met any of the following criteria: clinically significant (per investigator); accompanied by clinical symptoms; resulted in a change in study treatment; or required a change in concomitant therapy.
Time Frame: Assessed at each study visit from Baseline until 28 days after the last dose of study treatment (up to 36 weeks)
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) | Arm B: Faricimab, 1.5 mg Q4W | Arm C: Faricimab, 6 mg Q4W | Arm D: Faricimab, 6 mg Every 4-8 Weeks | Arm E: Ranibizumab 0.5 mg + Faricimab 6 mg Q4W
Number analyzed (Participants) | 67 | 46 | 39 | 46 | 64
Participants
  Low: number analyzed (Participants) | 46 | 32 | 22 | 30 | 44
  Low | 28 | 19 | 14 | 25 | 29
  High: number analyzed (Participants) | 67 | 46 | 39 | 45 | 64
  High | 4 | 1 | 1 | 2 | 6

28. Secondary Outcome: Number of Participants With Marked Laboratory Abnormalities in Hematology and Coagulation Tests, in All Participants
Description: Clinical laboratory tests for hematology and coagulation parameters were performed and any marked abnormal values (High or Low) were based on Roche's predefined standard reference ranges. Marked laboratory abnormalities are presented according to COG3007 abnormality criteria: Single, Not Last = abnormality detected at a single assessment, but not at the last assessment; Last or Replicated = abnormality detected at the last assessment or replicated at one or more assessments. Not every laboratory abnormality qualified as an adverse event, only if it met any of the following criteria: clinically significant (per investigator); accompanied by clinical symptoms; resulted in a change in study treatment; or required a change in concomitant therapy. Abs. = absolute count; Corp. = corpuscular; Ery. = erythrocyte; INR = International Normalized Ratio
Time Frame: Predose at Baseline, Weeks 12 and 36, and at Early Termination and Unscheduled Visits (up to 36 weeks)
Population: Safety Population: all participants who received at least one dose of study treatment. This analysis included participants with non-missing assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) | Arm B: Faricimab, 1.5 mg Q4W | Arm C: Faricimab, 6 mg Q4W | Arm D: Faricimab, 6 mg Every 4-8 Weeks | Arm E: Ranibizumab 0.5 mg + Faricimab 6 mg Q4W
Number analyzed (Participants) | 67 | 46 | 39 | 46 | 64
Participants
  Basophils, Abs., High - Any Abnormality: number analyzed (Participants) | 61 | 40 | 33 | 43 | 57
  Basophils, Abs., High - Any Abnormality | 1 | 0 | 0 | 0 | 0
  Basophils, Abs., High - Single, Not Last: number analyzed (Participants) | 61 | 40 | 33 | 43 | 57
  Basophils, Abs., High - Single, Not Last | 1 | 0 | 0 | 0 | 0
  Basophils, Abs., High - Last or Replicated: number analyzed (Participants) | 61 | 40 | 33 | 43 | 57
  Basophils, Abs., High - Last or Replicated | 0 | 0 | 0 | 0 | 0
  Eosinophils, Abs., High - Any Abnormality: number analyzed (Participants) | 61 | 40 | 35 | 43 | 58
  Eosinophils, Abs., High - Any Abnormality | 0 | 0 | 0 | 3 | 0
  Eosinophils, Abs., High - Single, Not Last: number analyzed (Participants) | 61 | 40 | 35 | 43 | 58
  Eosinophils, Abs., High - Single, Not Last | 0 | 0 | 0 | 1 | 0
  Eosinophils, Abs., High - Last or Replicated: number analyzed (Participants) | 61 | 40 | 35 | 43 | 58
  Eosinophils, Abs., High - Last or Replicated | 0 | 0 | 0 | 2 | 0
  Ery. Mean Corp. Volume, Low - Any Abnormality: number analyzed (Participants) | 65 | 43 | 38 | 44 | 62
  Ery. Mean Corp. Volume, Low - Any Abnormality | 0 | 0 | 0 | 1 | 0
  Ery. Mean Corp. Volume, Low - Single, Not Last: number analyzed (Participants) | 65 | 43 | 38 | 44 | 62
  Ery. Mean Corp. Volume, Low - Single, Not Last | 0 | 0 | 0 | 1 | 0
  Ery. Mean Corp. Volume, Low - Last or Replicated: number analyzed (Participants) | 65 | 43 | 38 | 44 | 62
  Ery. Mean Corp. Volume, Low - Last or Replicated | 0 | 0 | 0 | 0 | 0
  Hematocrit, Low - Any Abnormality: number analyzed (Participants) | 65 | 43 | 38 | 44 | 62
  Hematocrit, Low - Any Abnormality | 1 | 0 | 1 | 0 | 0
  Hematocrit, Low - Single, Not Last: number analyzed (Participants) | 65 | 43 | 38 | 44 | 62
  Hematocrit, Low - Single, Not Last | 1 | 0 | 1 | 0 | 0
  Hematocrit, Low - Last or Replicated: number analyzed (Participants) | 65 | 43 | 38 | 44 | 62
  Hematocrit, Low - Last or Replicated | 0 | 0 | 0 | 0 | 0
  Hemoglobin, Low - Any Abnormality: number analyzed (Participants) | 65 | 43 | 38 | 44 | 62
  Hemoglobin, Low - Any Abnormality | 3 | 0 | 1 | 2 | 2
  Hemoglobin, Low - Single, Not Last: number analyzed (Participants) | 65 | 43 | 38 | 44 | 62
  Hemoglobin, Low - Single, Not Last | 2 | 0 | 0 | 0 | 1
  Hemoglobin, Low - Last or Replicated: number analyzed (Participants) | 65 | 43 | 38 | 44 | 62
  Hemoglobin, Low - Last or Replicated | 1 | 0 | 1 | 2 | 1
  Lymphocytes, Abs., Low - Any Abnormality: number analyzed (Participants) | 55 | 39 | 34 | 42 | 54
  Lymphocytes, Abs., Low - Any Abnormality | 0 | 1 | 1 | 2 | 1
  Lymphocytes, Abs., Low - Single, Not Last: number analyzed (Participants) | 55 | 39 | 34 | 42 | 54
  Lymphocytes, Abs., Low - Single, Not Last | 0 | 1 | 1 | 0 | 1
  Lymphocytes, Abs., Low - Last or Replicated: number analyzed (Participants) | 55 | 39 | 34 | 42 | 54
  Lymphocytes, Abs., Low - Last or Replicated | 0 | 0 | 0 | 2 | 0
  Lymphocytes, Abs., High - Any Abnormality: number analyzed (Participants) | 55 | 39 | 34 | 42 | 54
  Lymphocytes, Abs., High - Any Abnormality | 0 | 0 | 0 | 1 | 0
  Lymphocytes, Abs., High - Single, Not Last: number analyzed (Participants) | 55 | 39 | 34 | 42 | 54
  Lymphocytes, Abs., High - Single, Not Last | 0 | 0 | 0 | 0 | 0
  Lymphocytes, Abs., High - Last or Replicated: number analyzed (Participants) | 55 | 39 | 34 | 42 | 54
  Lymphocytes, Abs., High - Last or Replicated | 0 | 0 | 0 | 1 | 0
  Lymphocytes, Pct., Low - Any Abnormality: number analyzed (Participants) | 10 | 4 | 4 | 2 | 8
  Lymphocytes, Pct., Low - Any Abnormality | 0 | 1 | 0 | 0 | 0
  Lymphocytes, Pct., Low - Single, Not Last: number analyzed (Participants) | 10 | 4 | 4 | 2 | 8
  Lymphocytes, Pct., Low - Single, Not Last | 0 | 1 | 0 | 0 | 0
  Lymphocytes, Pct., Low - Last or Replicated: number analyzed (Participants) | 10 | 4 | 4 | 2 | 8
  Lymphocytes, Pct., Low - Last or Replicated | 0 | 0 | 0 | 0 | 0
  Neutrophils, Total, Abs., Low - Any Abnormality: number analyzed (Participants) | 61 | 40 | 33 | 43 | 57
  Neutrophils, Total, Abs., Low - Any Abnormality | 0 | 1 | 2 | 3 | 1
  Neutrophils, Total, Abs., Low - Single, Not Last: number analyzed (Participants) | 61 | 40 | 33 | 43 | 57
  Neutrophils, Total, Abs., Low - Single, Not Last | 0 | 1 | 1 | 1 | 0
  Neutrophils, Total, Abs., Low - Last or Replicated: number analyzed (Participants) | 61 | 40 | 33 | 43 | 57
  Neutrophils, Total, Abs., Low - Last or Replicated | 0 | 0 | 1 | 2 | 1
  Neutrophils, Total, Abs., High - Any Abnormality: number analyzed (Participants) | 61 | 40 | 33 | 43 | 57
  Neutrophils, Total, Abs., High - Any Abnormality | 2 | 1 | 0 | 0 | 2
  Neutrophils, Total, Abs., High - Single, Not Last: number analyzed (Participants) | 61 | 40 | 33 | 43 | 57
  Neutrophils, Total, Abs., High - Single, Not Last | 1 | 0 | 0 | 0 | 2
  Neutrophils, Total, Abs., High -Last or Replicated: number analyzed (Participants) | 61 | 40 | 33 | 43 | 57
  Neutrophils, Total, Abs., High -Last or Replicated | 1 | 1 | 0 | 0 | 0
  Platelets, Low - Any Abnormality: number analyzed (Participants) | 65 | 43 | 38 | 44 | 62
  Platelets, Low - Any Abnormality | 0 | 0 | 0 | 2 | 1
  Platelets, Low - Single, Not Last: number analyzed (Participants) | 65 | 43 | 38 | 44 | 62
  Platelets, Low - Single, Not Last | 0 | 0 | 0 | 1 | 0
  Platelets, Low - Last or Replicated: number analyzed (Participants) | 65 | 43 | 38 | 44 | 62
  Platelets, Low - Last or Replicated | 0 | 0 | 0 | 1 | 1
  White Blood Cell Count, Low - Any Abnormality: number analyzed (Participants) | 65 | 43 | 38 | 44 | 62
  White Blood Cell Count, Low - Any Abnormality | 0 | 0 | 0 | 1 | 1
  White Blood Cell Count, Low - Single, Not Last: number analyzed (Participants) | 65 | 43 | 38 | 44 | 62
  White Blood Cell Count, Low - Single, Not Last | 0 | 0 | 0 | 1 | 1
  White Blood Cell Count, Low - Last or Replicated: number analyzed (Participants) | 65 | 43 | 38 | 44 | 62
  White Blood Cell Count, Low - Last or Replicated | 0 | 0 | 0 | 0 | 0
  White Blood Cell Count, High - Any Abnormality: number analyzed (Participants) | 65 | 43 | 38 | 44 | 62
  White Blood Cell Count, High - Any Abnormality | 0 | 0 | 0 | 1 | 0
  White Blood Cell Count, High - Single, Not Last: number analyzed (Participants) | 65 | 43 | 38 | 44 | 62
  White Blood Cell Count, High - Single, Not Last | 0 | 0 | 0 | 0 | 0
  White Blood Cell Count, High - Last or Replicated: number analyzed (Participants) | 65 | 43 | 38 | 44 | 62
  White Blood Cell Count, High - Last or Replicated | 0 | 0 | 0 | 1 | 0
  INR, High - Any Abnormality: number analyzed (Participants) | 2 | 2 | 1 | 3 | 1
  INR, High - Any Abnormality | 0 | 0 | 0 | 1 | 0
  INR, High - Single, Not Last: number analyzed (Participants) | 2 | 2 | 1 | 3 | 1
  INR, High - Single, Not Last | 0 | 0 | 0 | 0 | 0
  INR, High - Last or Replicated: number analyzed (Participants) | 2 | 2 | 1 | 3 | 1
  INR, High - Last or Replicated | 0 | 0 | 0 | 1 | 0

29. Secondary Outcome: Number of Participants With Marked Laboratory Abnormalities in Blood Chemistry Tests, in All Participants
Description: Clinical laboratory tests for blood chemistry parameters were performed and any marked abnormal values (High or Low) were based on Roche's predefined standard reference ranges. Marked laboratory abnormalities are presented according to COG3007 abnormality criteria: Single, Not Last = abnormality detected at a single assessment, but not at the last assessment; Last or Replicated = abnormality detected at the last assessment or replicated at one or more assessments. Not every laboratory abnormality qualified as an adverse event, only if it met any of the following criteria: clinically significant (per investigator); accompanied by clinical symptoms; resulted in a change in study treatment; or required a change in concomitant therapy. GGT = gamma-glutamyltransferase; SGOT/AST = serum glutamic oxaloacetic transaminase / aspartate aminotransferase; SGPT/ALT = serum glutamic pyruvic transaminase / alanine aminotransferase
Time Frame: Predose at Baseline, Weeks 12 and 36, and at Early Termination and Unscheduled Visits (up to 36 weeks)
Population: as for outcome 28
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) | Arm B: Faricimab, 1.5 mg Q4W | Arm C: Faricimab, 6 mg Q4W | Arm D: Faricimab, 6 mg Every 4-8 Weeks | Arm E: Ranibizumab 0.5 mg + Faricimab 6 mg Q4W
Number analyzed (Participants) | 67 | 46 | 39 | 46 | 64
Participants
  Alkaline Phosphatase, High - Any Abnormality: number analyzed (Participants) | 65 | 43 | 39 | 45 | 63
  Alkaline Phosphatase, High - Any Abnormality | 0 | 0 | 1 | 0 | 0
  Alkaline Phosphatase, High - Single, Not Last: number analyzed (Participants) | 65 | 43 | 39 | 45 | 63
  Alkaline Phosphatase, High - Single, Not Last | 0 | 0 | 1 | 0 | 0
  Alkaline Phosphatase, High - Last or Replicated: number analyzed (Participants) | 65 | 43 | 39 | 45 | 63
  Alkaline Phosphatase, High - Last or Replicated | 0 | 0 | 0 | 0 | 0
  Bicarbonate (CO2), Low - Any Abnormality: number analyzed (Participants) | 63 | 43 | 39 | 44 | 64
  Bicarbonate (CO2), Low - Any Abnormality | 1 | 1 | 0 | 1 | 1
  Bicarbonate (CO2), Low - Single, Not Last: number analyzed (Participants) | 63 | 43 | 39 | 44 | 64
  Bicarbonate (CO2), Low - Single, Not Last | 0 | 0 | 0 | 1 | 0
  Bicarbonate (CO2), Low - Last or Replicated: number analyzed (Participants) | 63 | 43 | 39 | 44 | 64
  Bicarbonate (CO2), Low - Last or Replicated | 1 | 1 | 0 | 0 | 1
  Bicarbonate (CO2), High - Any Abnormality: number analyzed (Participants) | 63 | 43 | 39 | 44 | 64
  Bicarbonate (CO2), High - Any Abnormality | 5 | 3 | 1 | 3 | 4
  Bicarbonate (CO2), High - Single, Not Last: number analyzed (Participants) | 63 | 43 | 39 | 44 | 64
  Bicarbonate (CO2), High - Single, Not Last | 3 | 0 | 1 | 0 | 2
  Bicarbonate (CO2), High - Last or Replicated: number analyzed (Participants) | 63 | 43 | 39 | 44 | 64
  Bicarbonate (CO2), High - Last or Replicated | 2 | 3 | 0 | 3 | 2
  Calcium, Low - Any Abnormality: number analyzed (Participants) | 65 | 43 | 39 | 45 | 64
  Calcium, Low - Any Abnormality | 0 | 1 | 0 | 0 | 0
  Calcium, Low - Single, Not Last: number analyzed (Participants) | 65 | 43 | 39 | 45 | 64
  Calcium, Low - Single, Not Last | 0 | 0 | 0 | 0 | 0
  Calcium, Low - Last or Replicated: number analyzed (Participants) | 65 | 43 | 39 | 45 | 64
  Calcium, Low - Last or Replicated | 0 | 1 | 0 | 0 | 0
  Calcium, High - Any Abnormality: number analyzed (Participants) | 65 | 43 | 39 | 45 | 64
  Calcium, High - Any Abnormality | 0 | 0 | 0 | 0 | 1
  Calcium, High - Single, Not Last: number analyzed (Participants) | 65 | 43 | 39 | 45 | 64
  Calcium, High - Single, Not Last | 0 | 0 | 0 | 0 | 1
  Calcium, High - Last or Replicated: number analyzed (Participants) | 65 | 43 | 39 | 45 | 64
  Calcium, High - Last or Replicated | 0 | 0 | 0 | 0 | 0
  Chloride, Low - Any Abnormality: number analyzed (Participants) | 65 | 43 | 39 | 45 | 64
  Chloride, Low - Any Abnormality | 1 | 1 | 0 | 0 | 2
  Chloride, Low - Single, Not Last: number analyzed (Participants) | 65 | 43 | 39 | 45 | 64
  Chloride, Low - Single, Not Last | 1 | 1 | 0 | 0 | 0
  Chloride, Low - Last or Replicated: number analyzed (Participants) | 65 | 43 | 39 | 45 | 64
  Chloride, Low - Last or Replicated | 0 | 0 | 0 | 0 | 2
  Creatine Kinase, High - Any Abnormality: number analyzed (Participants) | 64 | 43 | 38 | 44 | 62
  Creatine Kinase, High - Any Abnormality | 2 | 0 | 1 | 3 | 2
  Creatine Kinase, High - Single, Not Last: number analyzed (Participants) | 64 | 43 | 38 | 44 | 62
  Creatine Kinase, High - Single, Not Last | 0 | 0 | 0 | 1 | 1
  Creatine Kinase, High - Last or Replicated: number analyzed (Participants) | 64 | 43 | 38 | 44 | 62
  Creatine Kinase, High - Last or Replicated | 2 | 0 | 1 | 2 | 1
  Creatinine, High - Any Abnormality: number analyzed (Participants) | 65 | 43 | 39 | 45 | 64
  Creatinine, High - Any Abnormality | 0 | 1 | 0 | 0 | 0
  Creatinine, High - Single, Not Last: number analyzed (Participants) | 65 | 43 | 39 | 45 | 64
  Creatinine, High - Single, Not Last | 0 | 1 | 0 | 0 | 0
  Creatinine, High - Last or Replicated: number analyzed (Participants) | 65 | 43 | 39 | 45 | 64
  Creatinine, High - Last or Replicated | 0 | 0 | 0 | 0 | 0
  GGT, High - Any Abnormality: number analyzed (Participants) | 64 | 43 | 39 | 45 | 63
  GGT, High - Any Abnormality | 0 | 0 | 0 | 1 | 1
  GGT, High - Single, Not Last: number analyzed (Participants) | 64 | 43 | 39 | 45 | 63
  GGT, High - Single, Not Last | 0 | 0 | 0 | 0 | 0
  GGT, High - Last or Replicated: number analyzed (Participants) | 65 | 43 | 39 | 45 | 63
  GGT, High - Last or Replicated | 0 | 0 | 0 | 1 | 1
  Phosphorus, Low - Any Abnormality: number analyzed (Participants) | 62 | 42 | 37 | 44 | 61
  Phosphorus, Low - Any Abnormality | 0 | 1 | 1 | 0 | 1
  Phosphorus, Low - Single, Not Last: number analyzed (Participants) | 62 | 42 | 37 | 44 | 61
  Phosphorus, Low - Single, Not Last | 0 | 1 | 0 | 0 | 0
  Phosphorus, Low - Last or Replicated: number analyzed (Participants) | 62 | 42 | 37 | 44 | 61
  Phosphorus, Low - Last or Replicated | 0 | 0 | 1 | 0 | 1
  Phosphorus, High - Any Abnormality: number analyzed (Participants) | 62 | 42 | 37 | 44 | 61
  Phosphorus, High - Any Abnormality | 2 | 3 | 2 | 1 | 5
  Phosphorus, High - Single, Not Last: number analyzed (Participants) | 62 | 42 | 37 | 44 | 61
  Phosphorus, High - Single, Not Last | 1 | 1 | 1 | 1 | 3
  Phosphorus, High - Last or Replicated: number analyzed (Participants) | 62 | 42 | 37 | 44 | 61
  Phosphorus, High - Last or Replicated | 1 | 2 | 1 | 0 | 2
  Potassium, High - Any Abnormality: number analyzed (Participants) | 65 | 43 | 39 | 45 | 64
  Potassium, High - Any Abnormality | 2 | 1 | 0 | 0 | 1
  Potassium, High - Single, Not Last: number analyzed (Participants) | 65 | 43 | 39 | 45 | 64
  Potassium, High - Single, Not Last | 1 | 0 | 0 | 0 | 0
  Potassium, High - Last or Replicated: number analyzed (Participants) | 65 | 43 | 39 | 45 | 64
  Potassium, High - Last or Replicated | 1 | 1 | 0 | 0 | 1
  Protein, Total, High - Any Abnormality: number analyzed (Participants) | 65 | 43 | 39 | 45 | 63
  Protein, Total, High - Any Abnormality | 0 | 1 | 0 | 0 | 0
  Protein, Total, High - Single, Not Last: number analyzed (Participants) | 65 | 43 | 39 | 45 | 63
  Protein, Total, High - Single, Not Last | 0 | 1 | 0 | 0 | 0
  Protein, Total, High - Last or Replicated: number analyzed (Participants) | 65 | 43 | 39 | 45 | 63
  Protein, Total, High - Last or Replicated | 0 | 0 | 0 | 0 | 0
  SGOT/AST, High - Any Abnormality: number analyzed (Participants) | 65 | 43 | 39 | 45 | 63
  SGOT/AST, High - Any Abnormality | 0 | 0 | 1 | 0 | 1
  SGOT/AST, High - Single, Not Last: number analyzed (Participants) | 65 | 43 | 39 | 45 | 63
  SGOT/AST, High - Single, Not Last | 0 | 0 | 1 | 0 | 1
  SGOT/AST, High - Last or Replicated: number analyzed (Participants) | 65 | 43 | 39 | 45 | 63
  SGOT/AST, High - Last or Replicated | 0 | 0 | 0 | 0 | 0
  SGPT/ALT, High - Any Abnormality: number analyzed (Participants) | 65 | 43 | 39 | 45 | 63
  SGPT/ALT, High - Any Abnormality | 1 | 0 | 1 | 0 | 1
  SGPT/ALT, High - Single, Not Last: number analyzed (Participants) | 65 | 43 | 39 | 45 | 63
  SGPT/ALT, High - Single, Not Last | 0 | 0 | 1 | 0 | 1
  SGPT/ALT, High - Last or Replicated: number analyzed (Participants) | 65 | 43 | 39 | 45 | 63
  SGPT/ALT, High - Last or Replicated | 1 | 0 | 0 | 0 | 0

30. Secondary Outcome: Mean Change From Baseline in Intraocular Pressure in the Study Eye Over Time, in All Participants
Description: Intraocular pressure is the fluid pressure inside the eye. The method used to measure intraocular pressure (e.g., Goldmann tonometry) for each participant was to be applied consistently by the investigator throughout the study. On the day of dosing, intraocular pressure was monitored at 30 minutes post-treatment administration, and if intraocular pressure was ≥30 mmHg in the study eye, it was reassessed at 1 hour post-treatment administration.
Time Frame: Baseline, 0.5 hours postdose on Day 1, predose and 0.5 hours postdose at Weeks 4, 8, 12, 16, 20, 24, 28, and 32, and at Weeks 1, 13, and 36
Population: Safety Population: all participants who received at least one dose of study treatment
Measure: Mean (Standard Deviation); unit: millimetres of mercury (mmHg)
Arm/Group | Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) | Arm B: Faricimab, 1.5 mg Q4W | Arm C: Faricimab, 6 mg Q4W | Arm D: Faricimab, 6 mg Every 4-8 Weeks | Arm E: Ranibizumab 0.5 mg + Faricimab 6 mg Q4W
Number analyzed (Participants) | 67 | 46 | 39 | 46 | 64
millimetres of mercury (mmHg)
  Baseline (BL): Absolute Value | 15.07 (3.38) | 14.74 (3.08) | 14.69 (3.85) | 14.98 (2.91) | 14.27 (2.80)
  Change from BL at Day 1 (0.5 hr): number analyzed (Participants) | 67 | 45 | 39 | 46 | 63
  Change from BL at Day 1 (0.5 hr) | 1.90 (4.80) | 2.04 (5.32) | 1.59 (4.30) | 2.37 (4.22) | 3.52 (4.79)
  Change from BL at Week 1: number analyzed (Participants) | 65 | 46 | 39 | 46 | 64
  Change from BL at Week 1 | -0.89 (3.52) | -0.98 (3.47) | -0.62 (3.35) | -1.96 (2.98) | 0.11 (2.36)
  Change from BL at Week 4 (Predose): number analyzed (Participants) | 67 | 45 | 38 | 46 | 63
  Change from BL at Week 4 (Predose) | -0.27 (3.16) | -1.40 (2.61) | -1.18 (3.85) | -0.87 (2.99) | 0.59 (2.49)
  Change from BL at Week 4 (0.5 hr): number analyzed (Participants) | 67 | 44 | 37 | 45 | 61
  Change from BL at Week 4 (0.5 hr) | 2.88 (4.45) | 2.70 (3.56) | 2.05 (4.26) | 1.51 (3.96) | 3.59 (4.39)
  Change from BL at Week 8 (Predose): number analyzed (Participants) | 66 | 41 | 39 | 46 | 59
  Change from BL at Week 8 (Predose) | -0.56 (3.85) | -0.32 (3.13) | -0.69 (3.07) | -0.87 (2.75) | 0.10 (2.64)
  Change from BL at Week 8 (0.5 hr): number analyzed (Participants) | 66 | 41 | 38 | 46 | 58
  Change from BL at Week 8 (0.5 hr) | 2.70 (4.21) | 2.59 (4.64) | 2.37 (5.15) | 1.93 (3.91) | 3.93 (4.52)
  Change from BL at Week 12 (Predose): number analyzed (Participants) | 63 | 42 | 39 | 45 | 62
  Change from BL at Week 12 (Predose) | -0.17 (3.49) | -0.02 (2.88) | -0.82 (3.37) | 0.13 (2.94) | 0.45 (2.45)
  Change from BL at Week 12 (0.5 hr): number analyzed (Participants) | 62 | 42 | 37 | 45 | 61
  Change from BL at Week 12 (0.5 hr) | 3.08 (4.01) | 2.43 (3.41) | 2.59 (3.95) | 2.11 (4.04) | 4.34 (5.25)
  Change from BL at Week 13: number analyzed (Participants) | 61 | 40 | 38 | 43 | 57
  Change from BL at Week 13 | -0.77 (3.27) | -0.68 (3.12) | -0.71 (4.02) | -1.09 (2.70) | -0.65 (2.75)
  Change from BL at Week 16 (Predose): number analyzed (Participants) | 64 | 42 | 39 | 45 | 59
  Change from BL at Week 16 (Predose) | -0.41 (3.39) | 0.02 (3.10) | -0.77 (3.11) | -1.00 (2.56) | -0.36 (2.83)
  Change from BL at Week 16 (0.5 hr): number analyzed (Participants) | 64 | 41 | 39 | 43 | 59
  Change from BL at Week 16 (0.5 hr) | 1.64 (4.62) | 1.95 (5.35) | 1.67 (3.92) | -0.30 (3.98) | 3.12 (5.27)
  Change from BL at Week 20 (Predose): number analyzed (Participants) | 64 | 39 | 39 | 45 | 60
  Change from BL at Week 20 (Predose) | -0.16 (3.02) | -1.00 (2.73) | 0.08 (3.61) | -0.44 (3.18) | -0.17 (2.71)
  Change from BL at Week 20 (0.5 hr): number analyzed (Participants) | 64 | 39 | 39 | 44 | 60
  Change from BL at Week 20 (0.5 hr) | 2.80 (4.81) | 1.74 (4.85) | 1.82 (5.37) | 0.68 (5.45) | 2.62 (4.54)
  Change from BL at Week 24 (Predose): number analyzed (Participants) | 64 | 39 | 38 | 44 | 58
  Change from BL at Week 24 (Predose) | 0.00 (3.29) | -0.33 (3.30) | 0.26 (2.77) | -0.61 (2.73) | 0.14 (2.73)
  Change from BL at Week 24 (0.5 hr): number analyzed (Participants) | 64 | 39 | 35 | 44 | 58
  Change from BL at Week 24 (0.5 hr) | 3.23 (3.91) | 3.26 (4.04) | 4.11 (3.51) | 0.91 (3.66) | 4.17 (4.28)
  Change from BL at Week 28 (Predose): number analyzed (Participants) | 62 | 40 | 34 | 45 | 57
  Change from BL at Week 28 (Predose) | -0.02 (2.80) | 0.00 (4.30) | -1.00 (2.91) | -0.38 (2.74) | -0.19 (2.89)
  Change from BL at Week 28 (0.5 hr): number analyzed (Participants) | 62 | 39 | 34 | 45 | 57
  Change from BL at Week 28 (0.5 hr) | 3.16 (4.28) | 2.90 (4.13) | 1.74 (4.80) | 2.53 (3.60) | 3.86 (4.49)
  Change from BL at Week 32 (Predose): number analyzed (Participants) | 63 | 39 | 34 | 44 | 58
  Change from BL at Week 32 (Predose) | -0.73 (3.72) | -0.23 (3.63) | -0.41 (3.07) | -0.80 (2.92) | -0.67 (3.06)
  Change from BL at Week 32 (0.5 hr): number analyzed (Participants) | 62 | 39 | 32 | 43 | 57
  Change from BL at Week 32 (0.5 hr) | 1.81 (5.10) | 3.87 (5.58) | 1.63 (5.47) | -0.98 (4.38) | 2.37 (4.97)
  Change from BL at Week 36: number analyzed (Participants) | 64 | 40 | 37 | 44 | 58
  Change from BL at Week 36 | 0.00 (3.30) | 0.25 (3.68) | -0.65 (3.85) | -0.20 (3.55) | -0.16 (3.18)

31. Secondary Outcome: Change From Baseline in the Number of Participants With Anti-Drug Antibodies to Faricimab at Any Post-Baseline Timepoint
Description: Blood samples were obtained for measurement of anti-faricimab antibodies by a validated enzyme-linked immunosorbent assay (ELISA).
Time Frame: Baseline, Predose (0 hour) on Days 1, 28, 84, 112, 168, and 252 or early termination (up to 36 weeks)
Population: Safety Population: all participants who received at least one dose of study treatment. The analysis only included participants who received treatment with faricimab (i.e., Arm A was excluded) and had evaluable samples at baseline and any post-baseline timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) | Arm B: Faricimab, 1.5 mg Q4W | Arm C: Faricimab, 6 mg Q4W | Arm D: Faricimab, 6 mg Every 4-8 Weeks | Arm E: Ranibizumab 0.5 mg + Faricimab 6 mg Q4W
Number analyzed (Participants) | 0 | 46 | 38 | 46 | 63
Participants
  ADA Negative to Missing |  | 1 | 0 | 0 | 0
  ADA Negative to ADA Negative |  | 41 | 35 | 36 | 54
  ADA Negative to ADA Positive |  | 3 | 3 | 9 | 6
  ADA Positive to Missing |  | 0 | 0 | 0 | 0
  ADA Positive to ADA Negative |  | 1 | 0 | 0 | 0
  ADA Positive to ADA Positive |  | 0 | 0 | 1 | 3

32. Secondary Outcome: Mean Plasma Concentration of Faricimab Over Time, in All Participants
Description: Plasma concentrations of faricimab were measured by a specific validated enzyme-linked immunoabsorbent assay (ELISA) only from samples of participants randomized to receive faricimab. Baseline was defined as the last non-missing predose assessment. The lower limit of quantification (LLOQ) for the faricimab assay was 0.800 nanograms per millilitre (ng/mL). Values below the limit of quantification were imputed as LLOQ divided by 2.
Time Frame: Predose (on days when treatment was administered) at Baseline and Weeks 4, 12, 13, 16, 24, and 36
Population: Analysis included all randomized participants who had received treatment with faricimab (i.e., excludes Arm A at all timepoints and Arm E at Week 4) and had evaluable pharmacokinetic samples at a given timepoint.
Measure: Mean (Standard Deviation); unit: nanograms per millilitre (ng/mL)
Arm/Group | Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) | Arm B: Faricimab, 1.5 mg Q4W | Arm C: Faricimab, 6 mg Q4W | Arm D: Faricimab, 6 mg Every 4-8 Weeks | Arm E: Ranibizumab 0.5 mg + Faricimab 6 mg Q4W
Number analyzed (Participants) | 0 | 46 | 39 | 46 | 64
nanograms per millilitre (ng/mL)
  Baseline: number analyzed (Participants) | 0 | 46 | 39 | 45 | 63
  Baseline |  | 0.40 (0.00) | 0.40 (0.00) | 0.40 (0.00) | 0.47 (0.59)
  Week 4: number analyzed (Participants) | 0 | 45 | 38 | 44 | 0
  Week 4 |  | 8.83 (5.85) | 31.06 (18.47) | 36.58 (19.78) |
  Week 12: number analyzed (Participants) | 0 | 31 | 30 | 38 | 56
  Week 12 |  | 18.68 (24.38) | 57.92 (57.65) | 57.94 (73.91) | 45.29 (105.64)
  Week 13: number analyzed (Participants) | 0 | 46 | 39 | 46 | 62
  Week 13 |  | 43.32 (31.98) | 184.38 (102.01) | 178.25 (119.98) | 160.52 (124.73)
  Week 16: number analyzed (Participants) | 0 | 43 | 39 | 45 | 58
  Week 16 |  | 9.52 (7.41) | 46.99 (35.19) | 43.54 (39.05) | 44.71 (50.55)
  Week 24: number analyzed (Participants) | 0 | 39 | 38 | 45 | 58
  Week 24 |  | 9.07 (7.39) | 35.30 (22.03) | 31.19 (24.13) | 37.80 (27.75)
  Week 36: number analyzed (Participants) | 0 | 40 | 36 | 42 | 58
  Week 36 |  | 10.65 (8.47) | 36.43 (30.80) | 4.69 (7.24) | 36.06 (26.93)

33. Secondary Outcome: Mean Change From Baseline in Free Vascular Endothelial Growth Factor-A (VEGF-A) Plasma Concentrations Over Time, in All Participants
Description: The concentration of free VEGF was determined in plasma samples using an enzyme-linked immunosorbent assay (ELISA) method. The lower limit of quantification (LLOQ) of the assay was 15.6 picograms per millilitre (pg/mL). Plasma free VEGF concentrations below the limit of quantification were imputed as LLOQ divided by 2.
Time Frame: Baseline, Weeks 4, 12, 13, 16, 24, and 36
Population: Analysis included all randomized participants who had received study treatment and had evaluable pharmacodynamic samples at a given timepoint.
Measure: Mean (Standard Deviation); unit: picograms per millilitre (pg/mL)
Arm/Group | Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) | Arm B: Faricimab, 1.5 mg Q4W | Arm C: Faricimab, 6 mg Q4W | Arm D: Faricimab, 6 mg Every 4-8 Weeks | Arm E: Ranibizumab 0.5 mg + Faricimab 6 mg Q4W
Number analyzed (Participants) | 68 | 46 | 39 | 46 | 64
picograms per millilitre (pg/mL)
  Baseline (BL) - Value at Visit: number analyzed (Participants) | 64 | 46 | 39 | 43 | 61
  Baseline (BL) - Value at Visit | 15.25 (10.60) | 16.83 (12.08) | 24.63 (31.47) | 16.53 (9.73) | 22.60 (27.79)
  Change from BL at Week 4: number analyzed (Participants) | 61 | 45 | 38 | 40 | 60
  Change from BL at Week 4 | 0.52 (12.20) | 3.94 (33.25) | -9.26 (27.76) | -0.62 (15.67) | 3.75 (53.99)
  Change from BL at Week 12: number analyzed (Participants) | 50 | 33 | 32 | 35 | 52
  Change from BL at Week 12 | 1.52 (19.45) | -0.46 (13.30) | -8.58 (20.73) | -4.70 (11.79) | -3.24 (27.79)
  Change from BL at Week 13: number analyzed (Participants) | 52 | 27 | 27 | 31 | 37
  Change from BL at Week 13 | 2.62 (21.69) | 5.47 (52.19) | -14.10 (33.55) | -7.36 (10.67) | -15.14 (33.85)
  Change from BL at Week 16: number analyzed (Participants) | 60 | 39 | 38 | 40 | 54
  Change from BL at Week 16 | 12.12 (67.43) | -3.28 (10.61) | -9.86 (33.05) | -6.28 (10.84) | -5.34 (32.90)
  Change from BL at Week 24: number analyzed (Participants) | 60 | 38 | 38 | 40 | 53
  Change from BL at Week 24 | -0.67 (10.45) | 10.35 (50.09) | -12.57 (31.86) | -5.20 (10.07) | -7.19 (31.54)
  Change from BL at Week 36: number analyzed (Participants) | 57 | 40 | 36 | 36 | 55
  Change from BL at Week 36 | 1.91 (28.59) | -0.79 (11.86) | -12.16 (32.48) | -1.34 (13.69) | -8.17 (29.73)

34. Secondary Outcome: Mean Change From Baseline in Total Angiopoietin-2 (Ang-2) Plasma Concentrations Over Time, in All Participants
Description: Total Ang-2 concentrations were determined in plasma samples using an appropriate assay method. The lower limit of quantification (LLOQ) of the assay was 0.09 nanograms per millilitre (ng/mL). Plasma total Ang-2 concentrations below the limit of quantification were imputed as LLOQ divided by 2.
Time Frame: Baseline, Weeks 4, 12, 13, 16, 24, and 36
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: nanograms per millilitre (ng/mL)
Arm/Group | Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) | Arm B: Faricimab, 1.5 mg Q4W | Arm C: Faricimab, 6 mg Q4W | Arm D: Faricimab, 6 mg Every 4-8 Weeks | Arm E: Ranibizumab 0.5 mg + Faricimab 6 mg Q4W
Number analyzed (Participants) | 68 | 46 | 39 | 46 | 64
nanograms per millilitre (ng/mL)
  Baseline (BL) - Value at Visit: number analyzed (Participants) | 62 | 46 | 38 | 46 | 61
  Baseline (BL) - Value at Visit | 2.14 (1.38) | 1.81 (0.67) | 1.86 (1.12) | 1.80 (0.71) | 1.92 (0.95)
  Change from BL at Week 4: number analyzed (Participants) | 60 | 45 | 36 | 44 | 58
  Change from BL at Week 4 | 0.03 (0.48) | 0.09 (0.39) | 0.09 (0.27) | 0.20 (0.49) | -0.03 (0.38)
  Change from BL at Week 12: number analyzed (Participants) | 49 | 33 | 33 | 38 | 52
  Change from BL at Week 12 | 0.10 (0.89) | 0.14 (0.37) | 0.22 (0.48) | 0.19 (0.50) | -0.11 (0.49)
  Change from BL at Week 13: number analyzed (Participants) | 48 | 27 | 25 | 33 | 37
  Change from BL at Week 13 | 0.18 (0.91) | 0.23 (0.35) | 1.05 (1.15) | 0.87 (0.76) | 0.81 (0.98)
  Change from BL at Week 16: number analyzed (Participants) | 57 | 39 | 36 | 42 | 53
  Change from BL at Week 16 | 0.01 (0.62) | 0.04 (0.71) | 0.24 (0.47) | 0.22 (0.61) | -0.01 (0.52)
  Change from BL at Week 24: number analyzed (Participants) | 56 | 38 | 36 | 41 | 54
  Change from BL at Week 24 | 0.00 (0.68) | 0.11 (0.77) | 0.21 (0.52) | 0.24 (0.57) | 0.04 (0.44)
  Change from BL at Week 36: number analyzed (Participants) | 54 | 38 | 34 | 41 | 55
  Change from BL at Week 36 | 0.08 (0.42) | 0.05 (0.42) | 0.25 (0.39) | 0.33 (0.89) | 0.05 (0.56)

35. Secondary Outcome: Mean Change From Baseline in Free Angiopoietin-2 (Ang-2) Plasma Concentrations Over Time, in All Participants
Description: Free Ang-2 concentrations were determined in plasma samples using an appropriate assay method. The lower limit of quantification (LLOQ) of the assay was 0.9 nanograms per millilitre (ng/mL). Plasma free Ang-2 concentrations below the limit of quantification were imputed as LLOQ divided by 2.
Time Frame: Baseline, Weeks 4, 12, 13, 16, 24, and 36
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: nanograms per millilitre (ng/mL)
Arm/Group | Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) | Arm B: Faricimab, 1.5 mg Q4W | Arm C: Faricimab, 6 mg Q4W | Arm D: Faricimab, 6 mg Every 4-8 Weeks | Arm E: Ranibizumab 0.5 mg + Faricimab 6 mg Q4W
Number analyzed (Participants) | 68 | 46 | 39 | 46 | 64
nanograms per millilitre (ng/mL)
  Baseline (BL) - Value at Visit: number analyzed (Participants) | 62 | 46 | 38 | 46 | 61
  Baseline (BL) - Value at Visit | 2.19 (1.38) | 1.81 (0.73) | 1.88 (0.98) | 1.73 (0.75) | 1.95 (1.12)
  Change from BL at Week 4: number analyzed (Participants) | 60 | 45 | 36 | 44 | 58
  Change from BL at Week 4 | 0.00 (0.57) | 0.14 (0.37) | -0.05 (0.46) | 0.15 (0.62) | -0.07 (0.55)
  Change from BL at Week 12: number analyzed (Participants) | 49 | 33 | 33 | 38 | 53
  Change from BL at Week 12 | 0.23 (1.12) | 0.20 (0.57) | 0.12 (0.52) | 0.21 (0.75) | -0.01 (0.59)
  Change from BL at Week 13: number analyzed (Participants) | 48 | 27 | 25 | 33 | 37
  Change from BL at Week 13 | 0.03 (0.92) | 0.23 (0.69) | 0.81 (1.11) | 0.55 (0.75) | 0.32 (0.93)
  Change from BL at Week 16: number analyzed (Participants) | 57 | 39 | 37 | 42 | 53
  Change from BL at Week 16 | 0.06 (0.77) | 0.17 (0.95) | 0.15 (0.62) | 0.22 (0.67) | -0.11 (0.65)
  Change from BL at Week 24: number analyzed (Participants) | 56 | 38 | 36 | 41 | 54
  Change from BL at Week 24 | 0.18 (0.90) | 0.20 (0.93) | 0.25 (0.49) | 0.39 (0.58) | 0.13 (0.59)
  Change from BL at Week 36: number analyzed (Participants) | 54 | 38 | 34 | 41 | 55
  Change from BL at Week 36 | 0.16 (0.74) | 0.25 (0.65) | 0.28 (0.63) | 0.51 (1.30) | 0.06 (0.66)

ADVERSE EVENTS:
Time Frame: From Baseline until 28 days after the last dose of study treatment (up to 36 weeks)
Arm/Group | Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) | Arm B: Faricimab, 1.5 mg Q4W | Arm C: Faricimab, 6 mg Q4W | Arm D: Faricimab, 6 mg Every 4-8 Weeks | Arm E: Ranibizumab 0.5 mg + Faricimab 6 mg Q4W
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/46 | 0/39 | 0/46 | 1/64
Serious Adverse Events (participants affected / at risk) | 9/67 | 11/46 | 7/39 | 5/46 | 8/64
Other Adverse Events (participants affected / at risk) | 39/67 | 31/46 | 24/39 | 32/46 | 40/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) (N=67) | Arm B: Faricimab, 1.5 mg Q4W (N=46) | Arm C: Faricimab, 6 mg Q4W (N=39) | Arm D: Faricimab, 6 mg Every 4-8 Weeks (N=46) | Arm E: Ranibizumab 0.5 mg + Faricimab 6 mg Q4W (N=64)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cardiac disorder (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Degenerative mitral valve disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Glaucoma (Eye disorders) | 0 | 0 | 0 | 0 | 1
Keratic Precipitates (Eye disorders) | 0 | 1 | 0 | 0 | 0
Macular hole (Eye disorders) | 0 | 1 | 0 | 0 | 0
Neovascular age-related macular degeneration (Eye disorders) | 1 | 0 | 0 | 1 | 0
Retinal haemorrhage (Eye disorders) | 0 | 1 | 0 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Endophthalmitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Infectious colitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Arteriogram coronary (Investigations) | 0 | 0 | 1 | 0 | 0
Blood potassium increased (Investigations) | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Spindle cell sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pulmonary resection (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Shock (Vascular disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Ranibizumab, 0.5 mg Every 4 Weeks (Q4W) (N=67) | Arm B: Faricimab, 1.5 mg Q4W (N=46) | Arm C: Faricimab, 6 mg Q4W (N=39) | Arm D: Faricimab, 6 mg Every 4-8 Weeks (N=46) | Arm E: Ranibizumab 0.5 mg + Faricimab 6 mg Q4W (N=64)
Anterior chamber cell (Eye disorders) | 2 | 0 | 2 | 0 | 0
Blepharitis (Eye disorders) | 0 | 1 | 2 | 1 | 2
Cataract (Eye disorders) | 2 | 2 | 2 | 2 | 2
Conjunctival haemorrhage (Eye disorders) | 14 | 4 | 6 | 6 | 6
Dry age-related macular degeneration (Eye disorders) | 4 | 0 | 1 | 0 | 1
Eye irritation (Eye disorders) | 0 | 1 | 4 | 4 | 1
Eye pain (Eye disorders) | 2 | 4 | 2 | 5 | 3
Lacrimation increased (Eye disorders) | 1 | 0 | 1 | 3 | 0
Neovascular age-related macular degeneration (Eye disorders) | 6 | 4 | 3 | 2 | 5
Posterior capsule opacification (Eye disorders) | 2 | 1 | 3 | 0 | 1
Punctate keratitis (Eye disorders) | 0 | 0 | 0 | 0 | 5
Retinal pigment epithelial tear (Eye disorders) | 3 | 0 | 2 | 2 | 0
Vision blurred (Eye disorders) | 2 | 1 | 3 | 2 | 2
Vitreous detachment (Eye disorders) | 3 | 5 | 3 | 5 | 4
Vitreous floaters (Eye disorders) | 2 | 3 | 4 | 3 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 2 | 2 | 0 | 1
Influenza (Infections and infestations) | 3 | 3 | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 9 | 4 | 1 | 1 | 5
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 3 | 0
Urinary tract infection (Infections and infestations) | 6 | 11 | 2 | 0 | 3
Fall (Injury, poisoning and procedural complications) | 2 | 2 | 1 | 3 | 3
Intraocular pressure increased (Investigations) | 0 | 3 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 2 | 2 | 0
Weight increased (Investigations) | 0 | 0 | 2 | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 1 | 1 | 1 | 4
Insomnia (Psychiatric disorders) | 1 | 0 | 2 | 0 | 0
Hypertension (Vascular disorders) | 2 | 1 | 1 | 3 | 3
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 2
Anterior chamber flare (Eye disorders) | 3 | 1 | 0 | 0 | 1
Dry eye (Eye disorders) | 1 | 0 | 0 | 2 | 1
Visual acuity reduced (Eye disorders) | 1 | 1 | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 1 | 2 | 1
Pyrexia (General disorders) | 0 | 2 | 0 | 0 | 0
Sensation of foreign body (General disorders) | 0 | 1 | 0 | 2 | 0
Corneal abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 2
Cystitis (Infections and infestations) | 1 | 1 | 0 | 0 | 3
Gastroenteritis viral (Infections and infestations) | 3 | 0 | 0 | 1 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Sinusitis (Infections and infestations) | 2 | 1 | 0 | 1 | 2
Tooth abscess (Infections and infestations) | 1 | 2 | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 2 | 2
Red blood cell sedimentation rate increased (Investigations) | 0 | 0 | 1 | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 0 | 3
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 2 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 2
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 2 | 2
Headache (Nervous system disorders) | 0 | 2 | 0 | 2 | 2
Migraine (Nervous system disorders) | 0 | 2 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 2 | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 2 | 2

LIMITATIONS AND CAVEATS:
The small number of participants per cohort only allows detection of large differences in outcomes; not designed to show noninferiority of faricimab relative to ranibizumab. The short duration further limits information on long-term visual potential.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2016-09-09): https://cdn.clinicaltrials.gov/large-docs/90/NCT02484690/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-13): https://cdn.clinicaltrials.gov/large-docs/90/NCT02484690/SAP_001.pdf